

## NCT #NCT03761810

# Statistical Analysis Plan

Sol-Gel Technologies Ltd. SGT-65-05

Version: 2 Date: 26 NOV 2019

# STATISTICAL ANALYSIS PLAN

Protocol Number: SGT-65-05

Study Title: A Phase 3 Multi-Center, Double-Blind,

Randomized, Vehicle-Controlled Study of S6G5T-3 in the Treatment of Acne

Vulgaris

Development Phase of Study: 3

Sponsor: Sol-Gel Technologies Ltd.

Sponsor Contact:

Statistical Analysis Plan based on Protocol Version: 2.0

Statistical Analysis Plan Date:

26NOV2019

Statistical Analysis Plan Version: V2



Sol-Gel Technologies Ltd. SGT-65-05


SAP Approval

| - TI | |
|-------------------------------------|------------------|
| Authored by: | |
| SIGNATURE:QST Consultations, Ltd. | DATE: OZDECZO19 |
| Reviewed by: | |
| SIGNATURE: QST Consultations, Ltd. | DATE: 02DEC 2019 |
| Approved by: | |
| SIGNATURE: | DATE: |
| Sol-Gel Technologies Ltd. | |

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.




# SAP Change History

| Version | Date | Summary of Changes | Author |
|---|---|---|---|
| 1 | 02MAY2019 | Original document | |
| 2 | 26NOV2019 | In Section 8.1.11 an age grouping (9-11, 12-17 and 18-30, 31 and up) was added. | |
| | | In Section 8.7 the text was revised so that the secondary efficacy analysis is also being performed on the Per-Protocol population. | |
| | | In the table mocks the treatment header was updated to E-BPO/E-ATRA 3%/0.1% Cream for the active arm. | |
| | | In Section 8.4.4 the text ws updated to properly reflect the intended Week 12 window of +/- 4 days. | |




# TABLE OF CONTENTS

| 1. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | | | |
|---|---|---|---|---|
| 2. | PR | EFACE | | 8 |
| 3. | RE | SPONS | IBILITIES | 9 |
| 4. | INI | RODU | CTION | 9 |
| 5. | STU | J <b>DY O</b> I | BJECTIVES | 10 |
| | 5.1 | Prima | ry Objectives | 10 |
| | 5.2 | Secon | dary Objective | 11 |
| | 5.3 | Suppo | rtive Objective | 11 |
| | 5.4 | Safety | Objective | 11 |
| 6. | STU | STUDY DESIGN | | |
| | 6.1 | Overa | ll Study Design | 11 |
| | | 6.1.1 | Schedule of Visits and Assessments | 12 |
| | | 6.1.2 | Method of Assigning Subjects to Treatment Groups | 12 |
| | | 6.1.3 | Blinding | 13 |
| 7. | EFFICACY AND SAFETY ENDPOINTS | | | |
| | 7.1 | Efficacy Endpoints | | |
| | | 7.1.1 | Primary Efficacy Endpoints | 14 |
| | | 7.1.2 | Secondary Efficacy Endpoints | 14 |
| | | 7.1.3 | Supportive Efficacy Endpoints | 14 |
| | | 7.1.4 | Exploratory Endpoints | 15 |
| | 7.2 | Safety | Endpoints | 15 |
| 8. | STA | ATISTI | CAL AND ANALYTICAL PLANS | 15 |
| | 8.1 | | al Methodology | |
| | | 8.1.1 | Statistical Analysis | 16 |
| | | 8.1.2 | Baseline Definition | 16 |
| | | 8.1.3 | Visit Windowing | 16 |
| | | 8.1.4 | Adjustments for Covariates | 17 |
| | | 8.1.5 | Handling of Dropouts or Missing Data | 17 |
| | | | 8.1.5.1 Lesion Count Variable Missing Data Imputation | 18 |
| | | | 8.1.5.2 IGA Missing Data Imputation | |



Version: 2

Date: 26 NOV 2019

| | | 8.1.5.3 | PRE-FACE | Missing Data Imputation | 20 |
|---|---|---|---|---|---|
| | | 8.1.5.4 | Medication | Date Imputation | 21 |
| | 8.1.6 | Interim A | nalyses and Da | ata Monitoring | 21 |
| | 8.1.7 | Multicent | er Studies | | 21 |
| | 8.1.8 | Multiple Comparisons/Multiplicity | | | 24 |
| | 8.1.9 | Use of an | Efficacy Subs | et of Subjects | 24 |
| | 8.1.10 | Active-Co | ontrol Studies | Intended to Show Equivalence | 25 |
| | 8.1.11 | Examinat | ion of Subgrou | ıps | 25 |
| 8.2 | Dispos | ition of Sub | ojects | | 26 |
| 8.3 | Protoco | ol Deviation | ıs | | 26 |
| 8.4 | Data Se | ets Analyze | ed | | 26 |
| | 8.4.1 | Randomiz | zed Population | | 26 |
| | 8.4.2 | Intent-to- | Treat (ITT) Po | pulation | 27 |
| | 8.4.3 | Safety Pop | pulation | | 27 |
| | 8.4.4 | Per-Proto | col (PP) Popul | ation | 27 |
| 8.5 | Demog | raphic and | Other Baselin | e Characteristics | 28 |
| 8.6 | Prior an | nd Concom | itant Medicati | ons | 28 |
| 8.7 | Analys | is of Effica | cy | | 29 |
| | 8.7.1 | Primary E | Efficacy Analys | sis | 29 |
| | | 8.7.1.1 | Lesion Cour | nts | 29 |
| | | 8.7.1.2 | Investigator | Global Assessment (IGA) | 31 |
| | 8.7.2 | Sensitivity | y Efficacy Ana | ılysis | 31 |
| | | 8.7.2.1 | Sensitivity A | Analyses for Absolute Change in Lesion Count | 31 |
| | | | 8.7.2.1.1 | Repeated Measures | 31 |
| | | | 8.7.2.1.2 | Model Based Multiple Imputation | 31 |
| | | | 8.7.2.1.3 | Tipping Point | 32 |
| | | 8.7.2.2 | Sensitivity A | Analyses for IGA | 32 |
| | | | 8.7.2.2.1 | Repeated Measures | 32 |
| | | | 8.7.2.2.2 | Model Based Multiple Imputation | 33 |
| | | | 8.7.2.2.3 | Tipping Point | 33 |
| | 8.7.3 | Secondary | y Efficacy Ana | lysis | 34 |
| | 8.7.4 | Supportive Efficacy Analysis | | | 34 |
| | 8.7.5 | Explorato | ry Endpoint A | nalysis | 34 |
| 8.8 | Safety | Evaluation | | | 35 |
| | 8.8.1 | Extent of | Exposure | | 35 |



Version: 2

Date: 26 NOV 2019

| | 8.8.2 | Adverse 1 | Events (AEs) | 36 |
|-----|----------|------------|--------------------------------|-----|
| | 8.8.1 | Clinical I | Laboratory Evaluation | 37 |
| | 8.8.1 | Other Ob | oservations Related to Safety | 37 |
| | | 8.8.1.1 | Cutaneous Safety Assessments | |
| | | 8.8.1.2 | | |
| | | 8.8.1.3 | Vital Signs | |
| | | 8.8.1.4 | Physical Examination | 38 |
| | | | OF SAMPLE SIZEPLANNED ANALYSES | |
| 11. | REFEREN | CES | | 40 |
| 12. | INDEX OF | PLANNE | CD TABLES | 41 |
| 13. | INDEX OF | PLANNE | CD FIGURES | 172 |
| 14. | INDEX OF | PLANNE | CD LISTINGS | 174 |



Sol-Gel Technologies Ltd. SGT-65-05

Version: 2

Date: 26 NOV 2019

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

Acne-QoL Acne Quality-of-Life Questionnaire

AE(s) adverse event(s)

AID Acne impact domain

ANCOVA analysis of covariance

ANOVA analysis of variance

ATC Anatomical Therapeutic Chemical ASD acne sign and symptom domain

BMI body mass index

C Celsius

cm centimeters

CRF(s) case report form(s)

eCRF(s) electronic case report form(s)
E-BPO encapsulated benzoyl peroxide
FDA Food and Drug Administration

GCP good clinical practice

IGA Investigator Global Assessment

ITT Intent-to-Treat

IWRS Interactive Web Response System

kg kilograms

LOCF last observation carried forward

LSMean or LSM least square mean

max maximum

MCMC Markov Chain Monte Carlo

MedDRA Medical Dictionary for Regulatory Activities

mg milligram minimum

n number of observations

N number of subjects (sample size)

PRO Patient Reported Outcome

PRE-FACE Patient-Reported Evaluation of Facial Acne

PGI-C Patient Global Impression of Change



Sol-Gel Technologies Ltd. SGT-65-05

Version: 2

Date: 26 NOV 2019

| PGI-S | Patient Global Impression of Symptom Severity |
|--------|------------------------------------------------------|
| PGI-SE | Patient Global Impression of Treatments Side Effects |
| PGI-TS | Patient Global Impression of Treatments Satisfaction |

PP per-protocol PT preferred term

QST QST Consultations, Ltd. SAE(s) serious adverse event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

SD standard deviation SOC system organ class

TEAE(s) treatment-emergent adverse event(s)

WHO World Health Organization

#### 2. PREFACE

This Statistical Analysis Plan (SAP) describes the statistical analyses as it is foreseen before breaking the blind. The SAP will serve as a compliment to the study protocol and supersedes it in case of differences. In case of major differences between the study protocol and SAP, e.g. changes in the analysis related to the primary endpoint, a protocol amendment will be considered. The SAP may be updated during the study conduct and will be finalized before breaking the blind.

The following documents were reviewed in preparation of this SAP:

- Clinical Study Protocol SGT-65-05
  - Version 1.0 issued on 10OCT2018,
  - o Version 2.0 issued on 01NOV2018,
- Case report form (CRF) for SGT-65-05.
- ICH E9 Guidance on Statistical Principles for Clinical Trials.
- ICH E3 Structure and Content of Clinical Study Reports (CSRs)

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.



Sol-Gel Technologies Ltd. SGT-65-05


#### 3. RESPONSIBILITIES

The study statistician will be responsible for the statistical analysis planning. QST Consultations, Ltd. (QST), a Contract Research Organization (CRO) selected by Sol-Gel, will be responsible for the execution of all statistical programming deliverables. The statistical programming work will be supervised by the study statistician.

## 4. INTRODUCTION

Acne vulgaris is a common condition of the pilosebaceous units of the skin (hair follicles and oil glands). Acne is the most common skin disorder in the United States, affecting 40-50 million Americans. Acne usually begins in puberty, but the condition is not restricted to any age group.

Approximately 85% of people between the ages of 12 and 24 experience at least minor, most often on the face, chest, and back [1]. Acne is caused by four major factors:

- 1. Production of oil by enlarged oil glands in the skin.
- 2. Blockage of the hair follicles that release oil.
- 3. Growth of bacteria, called *Propionibacterium acnes*, within the hair follicles.
- 4. Inflammatory/immune response to *P. acnes*.

The pathophysiologic features of acne suggest that combination therapy should be utilized as early as possible to simultaneously attack the multiple pathogenic factors of the condition [2]. Antimicrobials have been a mainstay of acne treatment for many years, having multiple mechanisms of action. The most important may be the ability of antibiotics to decrease the number of *P. acnes* in and around the follicle. They have a bacteriostatic effect on *P. acnes*, which prevents the bacteria from producing pro-inflammatory molecules [3].

In June 2017, Sol Gel completed a double blind, randomized, dose ranging Phase 2 trial for S6G5T-3 involving 726 adult Patients at thirty-six centers in the United States (SGT-65-02: A Phase 2, Randomized, Double Blind, Active and Vehicle Controlled, 12-Week Study Evaluating the Efficacy, Safety, and Tolerability of S6G5T-3 and S6G5T-1 for the Treatment of Acne Vulgaris). The Phase 2 trial had two co primary endpoints: success in Investigator Global Assessment (IGA) namely, a two-grade reduction in IGA on a scale of 0 to 4 ("clear", "almost clear", "mild", "moderate", "severe") with "clear" or "almost clear" at Week 12; and a reduction in the mean inflammatory and non-inflammatory lesion count at Week 12 (end of trial). All Patients were 9 years of age or older with IGA of 3 or 4, 20 or more inflammatory lesions and 25 non-inflammatory lesions at enrollment. Patients were randomly divided into six groups of 119 to 122 Patients each and received a once daily dose, with one group receiving S6G5T-3 encapsulated benzoyl peroxide/encapsulated ATRA (E-BPO/E-ATRA 3%/0.1%), S6G5T-1

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Sol-Gel Technologies Ltd. SGT-65-05 Version: 2

Date: 26 NOV 2019

(E-BPO/E-ATRA (3%/0.05%), E-ATRA 0.1%, E-ATRA 0.05%, E-BPO 3% and Vehicle Cream alone. S6G5T-3 demonstrated numerical superiority to the active component E-BPO 3% and vehicle for the co-primary endpoints (treatment success and lesion counts inflammatory) at the Week 12 visit but only matched efficacy for non-inflammatory lesions for E-ATRA 0.1%. The success rate for at Least 2-Grade Improvement and Clear or Almost Clear was 12.27%, 22.10%, 31.72% and 39.68% for Vehicle Cream, E-BPO 3%, E-ATRA 0.1% and S6G5T-3, respectively. The mean inflammatory change from Baseline was -11.5, -13.8, -14.9 and -16.9. for Vehicle Cream, E-BPO 3%, E-ATRA 0.1% and S6G5T-3, respectively. The mean non-inflammatory change from Baseline was -13.7, -16.2, -23.8 and -23.6 for Vehicle Cream, E-BPO 3%, E-ATRA 0.1% and S6G5T-3, respectively. S6G5T-3 each demonstrated statistical superiority (p= 0.006 or less) to vehicle for the co-primary endpoints (treatment success, lesion counts both inflammatory and non-inflammatory) at the Week 12 visit.

In addition, S6G5T-3 were safe and well tolerated. The most common treatment-emergent adverse events (TEAEs) (≥5% incidence in any treatment group) were application site dryness, exfoliation and pain as well as upper respiratory infection. Cutaneous safety and tolerability assessment (erythema, scaling, pigmentation, itching, burning and stinging) by the Investigator showed that the proportion of Patients with these complaints tended to remain unchanged from Baseline over 12 weeks. On the other hand, based on self-assessments, a slightly greater proportion of Patients in the S6G5T-3 treatment groups had at least one higher post-baseline assessment of scaling, burning and stinging (mild) compared to vehicle. There were no apparent differences in mean changes from Baseline in any of the hematological and clinical chemistry test results in all treatment groups at Weeks 8 and 12. Most urinalysis test results were normal at Baseline and at Weeks 8 and 12. There were no clinically significant abnormalities in ECGs in the study.

In conclusion, both S6G5T-1 and S6G5T-3 demonstrate efficacy and safety in the treatment of acne vulgaris, however, S6G5T-3 showed additional benefit in achieving a greater proportion of treatment IGA success. Therefore, S6G5T-3 was selected as the "to be marketed formulation" and the active arm in this study.

#### 5. STUDY OBJECTIVES

# 5.1 Primary Objectives

The primary objectives of this pivotal study are:

• To assess the efficacy of S6G5T-3 compared to its Vehicle when applied once daily for 12 weeks in Patients with acne vulgaris.



Sol-Gel Technologies Ltd. SGT-65-05


• To assess the safety of S6G5T-3 when applied once daily for 12 weeks in Patients with acne vulgaris.

# 5.2 Secondary Objective

The secondary objective of this pivotal study is:

• To demonstrate statistical superiority in efficacy of Products S6G5T-3 as compared to the vehicle regarding percent change from Baseline.

# **5.3** Supportive Objective

The supportive objective of this pivotal study is:

• To determine the time required to observe improvement in the efficacy parameters associated with clearance of acne for Products S6G5T-3 compared to vehicle.

# 5.4 Safety Objective

The safety objectives of this pivotal study are:

• To determine the nature, severity and frequency of the adverse event (AE) rate and the localcutaneous reaction and tolerability of Products S6G5T-3 compared to the vehicle.

#### 6. STUDY DESIGN

# 6.1 Overall Study Design

This study will be a randomized, double-blind, multicenter, parallel group, active- and vehicle-controlled pivotal study to assess efficacy, and safety of Products S6G5T-3 and its vehicle for the treatment of acne vulgaris for 12 weeks. Approximately 420 Patients with moderate to severe acne vulgaris (rated 3 or 4 on the 5-point IGA) will be enrolled at up to 31 sites. Patients in this randomized, double-blind, vehicle-controlled, parallel-group multi-center study will be randomly assigned in a 2:1 ratio to Encapsulated Benzoyl Peroxide 3%/Encapsulated All-Trans-Retinoic Acids 0.1% (E-BPO/E-ATRA) Cream or Vehicle Cream respectively. Patients with severe acne vulgaris who are appropriate for systemic treatment need to be counseled regarding their treatment options by the Principal Investigator (PI).

The overall schedule of study visits includes:

- Visit 1/Screening
- Visit 2/Baseline, Day 1



Sol-Gel Technologies Ltd. SGT-65-05


- Visit 3/Week 2, Day 15 (± 3 Days)
- Visit 4/Week 4, Day 29 (± 3 Days)
- Visit 5/Week 8, Day 57 (± 3 Days)
- Visit 6/Week 12, Day 85 ( $\pm$  4 Days) / End of Study or Early Termination

Treatment efficacy will be evaluated using both clinician reported outcome (ClinRO) and Patient-reported outcome (PRO) questionnaires. Clinician reported efficacy assessments will include facial inflammatory and non-inflammatory lesion counts and an IGA which asks assessors to rate Patient's acne from 0 (Clear) to 4 (Severe). Patient reported efficacy assessments include the Patient-Reported Evaluation of Facial Acne (PRE-FACE), the Patient Global Impression of Symptom Severity (PGI-S), the Patient Global Impression of Change (PGI-C), and the Patient Global Impression of Treatments Satisfaction (PGI-TS).

Safety will be assessed at all visits and will include monitoring local and systemic AEs; the Investigator Cutaneous Safety Assessment rating of pigmentation, erythema, dryness and scaling on a scale ranging from 0 (None) to 3 (Severe) and the Patient assessment of Local Tolerability Assessment rating itching, burning and stinging on a scale ranging from 0 (None) to 3 (Severe). A Patient Global Impression of Treatment Side Effects (PGI-SE) will also be administered as part of the study design.

Clinician reported outcomes will be collected at study Visit 1, 2, 3, 4, 5 and 6. Patient-reported outcomes will be collected at study visit 2, 3, 4, 5, and 6 (with the exception of the PGI-C, PGI-TS and PGI-SE) which are not collected at Visit 1 or Visit 2). AEs and concomitant medications will be assessed throughout the treatment period. A urine pregnancy test is required at Visit 1, 2, 3, 4, 5 and 6 for all females of child-bearing potential and premenarchal.

#### 6.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 12.10 of the protocol.

# 6.1.2 Method of Assigning Subjects to Treatment Groups

It is planned that approximately 420 Patients, who meet the inclusion/exclusion criteria, will be enrolled in this study at up to 31 U.S. study sites. Patients will be at least 9 years of age and older, of either gender.

The study products will be administered in a double-blinded fashion (i.e., the treatment assignment will not be known to the Patient or to study personnel including Sol-Gel and its representatives). Patients will be instructed not to discuss the study product with the study personnel. Patients will be randomly assigned, in a 2:1 ratio, as follows:

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Sol-Gel Technologies Ltd. SGT-65-05


- E-BPO/E-ATRA 3%/0.1% Cream (Product S6G5T-3) (280 Patients)
- Vehicle Cream (Product S6G5T-8) (140 Patients)

Each Patient who signs an informed consent, meets inclusion/exclusion criteria, and successfully completes the screening procedures will be enrolled in the study. The Patient randomization schedule will be a permuted block design stratified by investigational site. Blocks will be composed of 3 treatment assignments in a ratio of 2:1 study product and vehicle respectively. Complete blocks from the randomization schedule will be allocated to investigational sites as they randomize Patients. Patients will be randomized through the IWRS and assigned a unique randomization ID assigning treatment group. The study product supplies will be packed in kits containing 4-pumps and will be numbered in a scrambled randomized method. The kits will be dispensed by the IWRS according to the Baseline assigned randomized treatment group.

# 6.1.3 Blinding

The staff involved in data management and statistical evaluation will remain blinded until identification of the analysis populations is completed and the database is locked.

The randomization schedule and treatment code will not be revealed to the Patients, study personnel, Sol-Gel or its representatives until after the database lock, except to the Medical Monitor or PI in the case of an emergency unblinding. Access to the randomization list will be maintained by and limited to the unblinded Biostatistician and the designated personnel directly responsible for labeling of study materials. The Medical Monitor will not have access to the randomization list, but may determine that unblinding of one or all Patients may be necessary in the case that the safety of study Patient(s) is at risk. In an emergency, the study blind may be broken only if:

- In the opinion of the Medical Monitor and/or the PI, it is in the Patient's best interest to do so.
- Knowledge of the treatment will alter the clinical management of the Patient.

In the case of an emergency that requires unblinding, the Investigator can request to unblind the Patient without prior contact with the Medical Monitor although follow-up between the Investigator and Medical Monitor must occur so that all parties are aware of the unblinding. Although it is recommended that the Investigator contact the Medical Monitor prior to unblinding any Patient, in instances where this is not feasible or advisable, the PI may directly access the Patient's treatment assignment. In all situations, the Interactive Web Response System (IWRS), will be used to obtain treatment assignment information, with limited access to only the



Sol-Gel Technologies Ltd. SGT-65-05


above-designated individuals; and any unblinding will be documented in the source records accordingly.

#### 7. EFFICACY AND SAFETY ENDPOINTS

# 7.1 Efficacy Endpoints

# 7.1.1 Primary Efficacy Endpoints

The co-primary efficacy endpoints are as follows:

- Proportion of Patients with an assessment of clear or almost clear and with at least a 2-grade improvement in IGA from Baseline at Week 12.
- Absolute change from Baseline in lesion count on the face at Week 12 (separately for inflammatory and non-inflammatory lesions).

# 7.1.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

- Percent change from Baseline, in non-inflammatory lesion count at Week 12.
- Percent change from Baseline, in inflammatory lesion count at Week 12.
- Proportion of Patients in the E-BPO/E-ATRA cream arm compared to vehicle control achieving at least a 4-point reduction on Item 1 (pimples) of the PRE-FACE from Baseline to Week 12.
- Proportion of Patients in the E-BPO/E-ATRA Cream arm compared to vehicle control achieving at least a 4-point reduction on Item 5 (embarrassment) of the PRE-FACE from Baseline to Week 12.
- Absolute change from Baseline, in non-inflammatory lesion count at Week 8
- Absolute change from Baseline, in inflammatory lesion count at Week 8.
- Absolute change from Baseline, in non-inflammatory lesion count at Week 4.
- Absolute change from Baseline, in inflammatory lesion count at Week 4.

# 7.1.3 Supportive Efficacy Endpoints

The supportive efficacy endpoints are as follows:



Sol-Gel Technologies Ltd. SGT-65-05


- Proportion of Patients with an assessment of clear or almost clear and with at least a 2-grade improvement in IGA from Baseline, at Weeks 2, 4 and 8.
- Absolute change from Baseline in inflammatory and non-inflammatory lesion counts from Baseline to Week 2.
- PRE-FACE ASD: Mean absolute change in PRE-FACE ASD scores from Baseline to Weeks 2, 4, and 8.
- PRE-FACE AID: Mean absolute change in PRE-FACE AID scores from Baseline to Weeks 2, 4, and 8.
- Proportion of Patients in treatment relative to control who report at least "minimally improved" as measured by the PGI-C at Week 12.
- Patient Global Impress of Symptom Severity (PGI-S) at Week 12.
- Patient Global Impression of Treatment Satisfaction (PGI-TS) at Week 12.

# 7.1.4 Exploratory Endpoints

The exploratory endpoint is the mean change in Acne-QoL domain scores from Baseline to Week 12.

# 7.2 Safety Endpoints

Safety will be assessed through Cutaneous Safety Assessment, Local Tolerability Assessment, AE reporting, physical examination, and vital signs.

## 8. STATISTICAL AND ANALYTICAL PLANS

## 8.1 General Methodology

All statistical processing will be performed using SAS® version 9.3 or later unless otherwise stated. Statistical significance will be based on two-tailed tests of the null hypothesis resulting in p-values of 0.05 or less.

The primary method of handling missing efficacy data will be based on estimation using the method of Markov Chain Monte Carlo (MCMC) imputation. The estimation will be done for each treatment group separately so that the pattern of missingness for one group does not influence the estimation of missing data for another group. Groups of complete datasets following the estimation will be concatenated to form analysis datasets for the comparative



Sol-Gel Technologies Ltd. SGT-65-05


analyses and subsequent imputation result inference with SAS PROC MIANALYZE. Descriptive statistics will also be derived from the multiply imputed datasets.

Sensitivity analyses for the primary efficacy endpoints will use 3 methods. For the lesion count endpoint, the first method will use a repeated measures analysis of covariance (ANCOVA), with treatment, analysis center, visit (i.e., Week 2, Week 4 and Week 8), and treatment group by visit interaction as independent factors and a covariate of Baseline. In this analysis, data from all post-baseline visits will be included with no imputation for missing data.

The second sensitivity analyses will use the model based multiple imputation method to impute missing data for the absolute change at Week 12.

The third sensitivity analysis will involve a tipping point analysis.

Similar methods for the dichotomized IGA will involve a repeated measures logistic regression model and a model based multiple imputation and tipping point analysis.

# 8.1.1 Statistical Analysis

All analyses will be performed by QST using SAS® Version 9.3 or later. All summary tables and data listings will be prepared utilizing SAS® software.

The standard operating procedures (SOPs) of QST will be followed in the creation and quality control of all data displays and analyses.

All data listings will be by subject. Additionally, all listings except the screen failure and randomization listings will be by treatment.

#### **8.1.2** Baseline Definition

Baseline is defined as the last non-missing assessment prior to first application of study drug. If the date of first application is unknown due to the subject being lost to follow-up, the Baseline visit record will be used as Baseline if it is non-missing. Missing results will not be flagged as Baseline.

# 8.1.3 Visit Windowing

Data will be summarized based on nominal visit indications with the exception of data captured at early termination and unscheduled visits. Data from early termination and unscheduled visits will be summarized based on mapped visit values. The analysis windows for early termination and unscheduled visits are presented in the following table.



Sol-Gel Technologies Ltd. SGT-65-05


# **Analysis Windows for Efficacy and Safety Assessments**

| Scheduled Visit | Target Study Day | Window (Days) |
|-----------------|------------------|---------------|
| Week 2 | 15 | 8 to 21 |
| Week 4 | 29 | 22 to 42 |
| Week 8 | 57 | 43 to 70 |
| Week 12 | 85 | 71 to 98 |

Data collected at early termination and unscheduled visits prior to study day 8 will not be analyzed, with the exception of those identified as Baseline values. Data collected at early termination and unscheduled visits after study day 98 will not be included in analyses.

The definition for the study day included in each study window is defined as below:

Study Day on or after Day 
$$1 = Visit Date - Day 1 Date + 1$$

If an assessment's mapped visit is a visit at which the subject has data from a scheduled visit present, or if no analyses are planned for the assessment at the mapped visit, the data collected at the early termination or unscheduled visit will not be included in analyses.

In the event of multiple values from unscheduled or early termination assessments within an analysis window, the value closest to the scheduled visit target study day will be used for analyses. If two values tie as closest to the time point (for example, one value is before and the other value is after the time point), then the later value will be selected.

Data collected at all visits will be included in the data listings with visit presented as reported by the site.

# 8.1.4 Adjustments for Covariates

Baseline lesion count will be a covariate for the primary efficacy endpoint for acne lesion counts. No other covariates are planned to be used in the analyses for this study.

# 8.1.5 Handling of Dropouts or Missing Data

Missing data for the ITT population will be estimated by multiple imputation and subsequently analyzed. Missing lesion count and IGA data will be derived for the analysis using the method of Markov Chain Monte Carlo (MCMC) multiple imputation. The pattern of missing observations



Sol-Gel Technologies Ltd. SGT-65-05


in each treatment group cannot influence the missing value estimation in the other group because the imputation will be conducted independently for each treatment group.

Last observation carried forward (LOCF) will be used to impute missing data for the efficacy analyses using the Per Protocol (PP) population.

Patients that discontinue from the study due to an AE related to study treatment or documented lack of treatment effect will be included in the PP population. Data for these subjects will not be imputed by multiple imputation or LOCF but rather their data will be imputed with values consistent with their status as treatment failures. For these subjects, values for lesion count and IGA will be imputed such that change from Baseline is zero, meaning the values will be set to the Baseline value. This imputation will be done after the data for all subjects has been through the MI process.

Incomplete start and end dates for medications will be imputed. Other safety data will not be imputed and will be summarized on an observed case basis.

# 8.1.5.1 Lesion Count Variable Missing Data Imputation

Multiple imputation and subsequent analysis will involve 3 distinct phases with these principal tasks:

1. Create a data set of patients, one for each treatment group, with observed values and those needing estimation by MCMC. The missing lesion count values in each data set will be filled in using the MCMC method 5 times to generate 5 data sets. The resulting data sets for each treatment arm will be combined into one complete data set for each imputation.

#### Syntax:

```
proc mi data=datain out=dataout seed=&seed. nimpute=5 <options>;
  where trtpn=(1, or 2);
  mcmc chain=multiple;
  var baseline week2 week4 week8 week12;
run;
```

- 2. For each complete data set, the variable of interest for Baseline minus the Week 12 value for the week imputed will be computed. Each complete data set will be analyzed as specified for the particular analysis.
- 3. The results from these analyses will be combined into a single inference using SAS PROC MIANALYZE.



Sol-Gel Technologies Ltd. SGT-65-05


A total of 4 random seeds are needed to impute lesion counts. The following 4 random seeds have been pre-specified by using a random number generator:

- Inflammatory Lesion Counts; S6G5T-3: Seed = 577660451
- Inflammatory Lesion Counts; S6G5T-8 Vehicle: Seed = 1077045427
- Non-inflammatory Lesion Counts; S6G5T-3: Seed = 2132522555
- Non-inflammatory Lesion Counts; S6G5T-8 Vehicle: Seed = 2096664573

# 8.1.5.2 IGA Missing Data Imputation

A similar procedure will be used for the analyses based on proportion of IGA successes wherein the ANCOVA analysis is replaced with a logistic regression analysis. Specifically, missing IGA values from which the dichotomized IGA is derived will be estimated by MCMC. The pattern of missing observations in each treatment group cannot influence the missing value estimation in the other because the imputation is being conducted independently for each treatment group.

The missing IGA values will be derived for the analysis using the method of MCMC multiple imputation. Multiple imputation and subsequent analysis will involve 3 principal tasks:

1. Create a data set, one for each treatment group, of patients with observed values and those needing estimation by MCMC. The missing IGA values in each data set will be filled in using the MCMC method 5 times to generate 5 data sets. The resulting data sets for each treatment arm will be combined into one complete data set by imputation.

#### Syntax:

```
proc mi data=datain out=dataout seed=&seed. nimpute=5 <options>;
  where trtpn=(1, or 2);
  mcmc chain=multiple;
  var baseline week2 week4 week8 week12;
run:
```

- 2. For each complete data set, the dichotomous success rate (clear or almost clear with a 2-point change from Baseline) will be computed. The estimated global values will be rounded to the nearest integer value prior to evaluating the success rate. Each complete data set will be analyzed with a logistic regression with factors of treatment group and analysis center.
- 3. The results from these analyses will be combined into a single inference using SAS PROC MIANALYZE.

The following 2 random seeds have been pre-specified by using a random number generator:



Sol-Gel Technologies Ltd. SGT-65-05


• IGA; S6G5T-3: Seed = 1024310713

• IGA; S6G5T-3 Vehicle: Seed = 1659491795

# 8.1.5.3 PRE-FACE Missing Data Imputation

The same procedure will be used for the analyses based on proportion of PRE-FACE item 1 (pimples) and item 5 (embarrassment) successes as the IGA success. Specifically, missing PRE-FACE items 1 and 5 values from which the dichotomized versions are derived will be estimated by MCMC. The pattern of missing observations in each treatment group cannot influence the missing value estimation in the other because the imputation is being conducted independently for each treatment group.

The missing PRE-FACE items 1 and 5 values will be derived for the analysis using the method of MCMC multiple imputation. Multiple imputation and subsequent analysis will involve 3 principal tasks:

1. Create a data set, one for each treatment group, of patients with observed values and those needing estimation by MCMC. The missing PRE-FACE items 1 and 5 values in each data set will be filled in using the MCMC method 5 times to generate 5 data sets. The resulting data sets for each treatment arm will be combined into one complete data set by imputation.

#### Syntax:

```
proc mi data=datain out=dataout seed=&seed. nimpute=5 <options>;
  where trtpn=(1, or 2);
  mcmc chain=multiple;
  var baseline week2 week4 week8 week12;
run;
```

- 2. For each complete data set, the dichotomous success rate (at least a 4-point reduction from Baseline) will be computed. The estimated global values will be rounded to the nearest integer value prior to evaluating the success rate. Each complete data set will be analyzed with a logistic regression with factors of treatment group and analysis center.
- 3. The results from these analyses will be combined into a single inference using SAS PROC MIANALYZE.

The following 4 random seeds have been pre-specified by using a random number generator:

- PRE-FACE Pimples Scores; S6G5T-3: Seed = 3965781
- PRE-FACE Pimples Scores; S6G5T-3 Vehicle: Seed = 96876327



Sol-Gel Technologies Ltd. SGT-65-05


- PRE-FACE Embarrassment Scores; S6G5T-3: Seed = 852215120
- PRE-FACE Embarrassment Scores; S6G5T-3 Vehicle: Seed = 1366717274

# **8.1.5.4 Medication Date Imputation**

If the medication start date is incomplete, then it will be imputed as follows for the purpose of determining concomitant use:

- If the start date is completely missing, the start date will be equal to the first dose date. However, if the stop date is not missing and is before the first dose date, then the stop date will be used instead.
- If the start day is missing, the first day of the month will be used.
- If the start day and month are missing, then the first day of the first month (January) will be used.

If the medication stop date is incomplete, then it will be imputed as follows for the purpose of determining concomitant use:

- If the stop date is completely missing and the medication is not ongoing, the stop date will be equal to the last dose date or date of completion/withdrawal, whichever is the latest.
- If the stop day is missing, the last day of the month will be used.

If the stop day and month are missing, then the last day of the last month (December) will be used.

# 8.1.6 Interim Analyses and Data Monitoring

No interim analysis or data monitoring is planned for this study.

#### 8.1.7 Multicenter Studies

The clinical study will be conducted under a common protocol for each investigational site with the intention of pooling the data for analysis. Every effort will be made to promote consistency in study execution at each investigational site. The study is intended to be conducted in a manner such that a minimum of 15 subjects will be randomized and included in the ITT population (i.e., at least ten subjects in the active treatment arm and five subjects in the vehicle treatment arm) for any investigator. In the event that there are too few subjects in a treatment arm for an



Sol-Gel Technologies Ltd. SGT-65-05 Version: 2

Date: 26 NOV 2019

investigational site, then the site's data will be combined with other site's data to achieve the desired sample size minimum per treatment arm. The combining of investigator data will be accomplished by taking the data of the investigator with the smallest enrollment and combining them with the data of the investigator with the largest enrollment, restricted to investigational sites which did not meet minimum enrollment. If there is a further need to combine data, then the data of the investigator with the second smallest enrollment will be combined with the site's data which had the second largest enrollment (restricted to investigational sites which did not meet minimum enrollment), and so on. This process will continue for all investigators who did not have a minimum of 15 subjects enrolled. The process of combining investigator data that have insufficient subjects per treatment arm will result in redefining the groups of investigators for the purposes of statistical analyses. These combined groups will be referred to as "analysis centers" in the statistical analyses.

The consistency of treatment response will be investigated across the analysis centers subsequent to combining the data as described above. Statistical tests will be conducted to identify if there are extreme analysis centers that could affect the interpretation of common statistical and clinical conclusions. An analysis center by treatment interaction will be included in the primary analyses to test for parallel treatment effect at an alpha level of 0.10. Change from Baseline in inflammatory and non-inflammatory lesions will be analyzed with an ANCOVA (unranked or ranked) with factors of treatment group, analysis center and treatment group by analysis center interaction and the respective Baseline lesion count variable as a covariate. For the purpose of testing consistency of treatment response, the dichotomized IGA will be analyzed with a logistic regression with factors of treatment group, analysis center, and the interaction term of treatment group by analysis center. Further examination will follow for any variables that have a significant ANCOVA or logistic regression interaction term.

In the event that the ANCOVA or logistic regression interaction (referred to henceforth as the "appropriate test") p-value is less than or equal to 0.10, a sensitivity analysis that excludes analysis centers with the extreme efficacy result will be performed to determine the robustness of the treatment effect. On the other hand, if all three analyses result in interaction terms with p-values greater than 0.10, then the conclusions from the pooled data will be considered to be free of the impact of extreme analysis centers.

The first step in conducting a sensitivity analysis is to identify the extreme analysis center or centers that contribute to the statistical significance of the appropriate test. The process involves submitting subsets of analysis centers to the appropriate test and observing the appropriate test p-value for the subset. Subsets with p-values greater than 0.10 for the appropriate test are considered homogeneous.



Sol-Gel Technologies Ltd. SGT-65-05 Version: 2

Date: 26 NOV 2019

The search for an extreme analysis center begins by analyzing all subsets that can be created by excluding one analysis center. If one or more of the subsets result in an appropriate test p-value greater than or equal to 0.10, then the analysis center excluded from the subset with the largest p-value for the appropriate test is deemed to be the extreme analysis center.

If all appropriate test subset p-values are less than or equal to 0.10, then the process will analyze the appropriate test for all subsets that can be created by excluding two analysis centers. If one or more of these subsets generate appropriate test p-values larger than 0.10, then the analysis centers excluded from the subset with the largest appropriate test p-value are deemed the extreme analysis centers.

Thus, the process of identifying the extreme analysis centers will continue in a stepwise manner by first excluding one, then two, then three, etc., analysis centers until the appropriate test p-value exceeds 0.10.

Once the extreme analysis center or centers have been identified, then the treatment p-values of the remaining analysis centers will be computed. Inferences will be drawn from the treatment p-value, as well as any pertinent observations regarding the extreme analysis center or centers. Additionally, it is noted that this process excludes patients from the analysis in a non-random manner and has an unpredictable impact on the power of the treatment effect test. In the event that the treatment effect of the remaining subset is not statistically significant, due consideration of the post-hoc aspects of the process will be given when the results are interpreted. Conclusions will be presented by the Sponsor as appropriate to the findings of the sensitivity analysis.

Prior to investigating the treatment effect within the analysis centers, the treatment effect within investigational site will be investigated to determine if the site-to-site variability is such that it could mask the analysis center effects. Thus, prior to pooling, change from Baseline in inflammatory and non-inflammatory lesions will be analyzed with an ANCOVA (unranked or ranked) with factors of treatment group, investigational site, and treatment group by investigational site interaction, and the respective Baseline lesion count variable as a covariate. The dichotomized primary endpoint will be analyzed with a logistic regression with factors of treatment group, investigational site, and the interaction term of treatment group by investigational site. If any of the analyses are not computationally feasible due to some investigational sites having very few subjects enrolled, the low-enrolling investigational sites will be excluded from the analysis.



Sol-Gel Technologies Ltd. SGT-65-05


# 8.1.8 Multiple Comparisons/Multiplicity

The overall Type I error will be controlled by requiring the three co-primary efficacy endpoints to be statistically significant. Specifically, failure of either one of the primary efficacy endpoints will invalidate the statistical significance of the secondary efficacy endpoints.

Evaluation of the secondary efficacy variables will use a gated sequential procedure starting with the comparisons of the first step and proceeding onto the next step and etc.

A stepwise process will be conducted for testing the secondary efficacy endpoints in order to control for multiplicity. These tests will be performed for only the ITT population. The testing process will terminate whenever a statistical test for a step is not significant. All subsequent tests for the remaining steps will be considered not significant. The order of testing is provided below.

| Step<br>Number | Secondary Endpoint |
|---|---|
| 1 | Percent change from Baseline, in non-inflammatory lesion count at Week 12. |
| 2 | Percent change from Baseline, in inflammatory lesion count at Week 12. |
| 3 | Proportion of patients in the E-BPO/E-ATRA cream arm compared to vehicle control achieving at least a 4-point reduction on Item 1 (pimples) of the PREFACE from Baseline to Week 12. |
| 4 | Proportion of patients in the E-BPO/E-ATRA Cream arm compared to vehicle control achieving at least a 4-point reduction on Item 5 (embarrassment) of the PRE-FACE from Baseline to Week 12. |
| 5 | Absolute change from Baseline, in non-inflammatory lesion count at Week 8 |
| 6 | Absolute change from Baseline, in inflammatory lesion count at Week 8. |
| 7 | Absolute change from Baseline, in non-inflammatory lesion count at Week 4 |

# 8.1.9 Use of an Efficacy Subset of Subjects

Subjects randomized to study drug who were dispensed study product and do not have major protocol deviations will form the PP Population. The requirements for the PP Population are outlined in Section 8.4.4. Any additional major protocol deviations will be defined at the time of evaluability evaluation, the time between the database soft lock and hard lock before unblinding.

Excluding subjects who have major protocol deviations will decrease the variability in treatment response and will allow for a better determination of dose-response relationship of S6G5T-3.



Sol-Gel Technologies Ltd. SGT-65-05


# 8.1.10 Active-Control Studies Intended to Show Equivalence

Not applicable to this study.

# **8.1.11** Examination of Subgroups

Subset analyses will be conducted for the ITT populations for the subgroups based on at least the following:

- Baseline Global Severity;
  - Categorized as Baseline IGA = 3 (moderate) and Baseline IGA = 4 (severe); due to the inclusion criteria requiring subjects to have either a 3 or 4 IGA score at study entry other IGA response categories will not be presented
- Sex;
  - Male versus female subjects
- Age;
  - Dichotomized to less than the median age of ITT subjects and greater than or equal to the median age of ITT subjects
  - Categories of less than 18,18 to less than the median age of ITT subjects and greater than or equal to the median age of ITT subjects; if the median age of ITT subjects is 18 or less, the subgroup will be less than 18 and greater than or equal to 18
  - o Categories of 9-11 years, 12-17 years, 18-30 years, and 31 years and older
- Ethnicity;
  - Categorized as Hispanic or Latino and Not Hispanic or Latino; ethnicities of Not Reported and Unknown will not be included
- Race
  - Categorized as White and Non-White; subjects indicating more than one race category which includes both white and a non-white race will be summarized under the Non-White subgroup.



Sol-Gel Technologies Ltd. SGT-65-05


Subset analyses will be conducted on the variables absolute change from Baseline in inflammatory lesions at Week 12 as well as the dichotomized global severity score at Week 12. These analyses will contain only descriptive statistics.

## 8.2 Disposition of Subjects

The number of subjects included in each analysis population (randomized, ITT, Safety, and PP) will be summarized by treatment group and overall. The number of subjects completed and discontinued (including the reasons for discontinuation) will be summarized for each treatment group as well as by overall. The percentages will be calculated based on the number of randomized patients, unless otherwise specified.

#### **8.3** Protocol Deviations

In order to define the PP Population, protocol deviations potentially influencing the evaluation of the primary efficacy endpoint will be defined as major deviations. The protocol deviations that will exclude a subject from PP are given in Section 8.4.4.

In case other deviations detected during the study conduct are considered to potentially influence the evaluation of the primary efficacy endpoint, these deviations will be documented prior to the database lock and the patients having these deviations will be excluded from the PP Population.

All protocol deviations will be reported to the sponsor and recorded throughout the study. Protocol deviations will not be entered into the database. SolGel will provide a list of protocol deviations to QST. A tabulation of protocol deviations will be presented in a data listing.

# 8.4 Data Sets Analyzed

Subjects will be presented/summarized based on the primary reason for exclusion. Below is the order to be used in summaries:

# **8.4.1** Randomized Population

All subjects who are randomized to study treatment will be included in the randomized population and will be analyzed according to the treatment group they were randomized. Listings will be provided for all randomized subjects.



Sol-Gel Technologies Ltd. SGT-65-05


# 8.4.2 Intent-to-Treat (ITT) Population

All subjects in the randomized population who are dispensed study product will be included in the ITT population and will be analyzed according to the treatment group they were randomized. All efficacy analyses will be presented using the ITT population.

# 8.4.3 Safety Population

All subjects in the randomized population who are presumed to have used the study product at least once and who provide at least one post-baseline safety evaluation will be included in the Safety population and will be analyzed according to the treatment they received. Presumed to have used study product will be defined as having at least one confirmed application of study medication. All safety analyses will be performed using the Safety population.

# 8.4.4 Per-Protocol (PP) Population

All subjects in the ITT population who complete the Week 12 evaluation without any significant protocol violations will be included in the PP population and analyzed according to the treatment group they received. The PP population will include subjects in the ITT population who do not meet any of the following criteria:

- Failed any of the inclusion/exclusion criteria;
- Have taken any interfering concomitant medications;
- Did not attend the Week 12 Visit;
- Missed more than 1 post-baseline study visit prior to Week 12;
- Have not been compliant with the dosing regimen (i.e., Patients may not miss more than five consecutive days of applications and must take 80-120% of expected applications. The number of expected applications will be determined for each Patient based on the length of their participation in the study);
- Out of visit window (+/- 4 days) at the 12-week Visit.

Subjects that discontinue from the study due to an AE related to study treatment or documented lack of treatment effect will be included in the PP population. Data for these subjects will not be imputed by multiple imputation but rather their data will be imputed with values consistent with their status as treatment failures. See Section 8.1.5 for additional detail. Prior to breaking the blind, other additional criteria may be added to the list to accommodate for unforeseen events that may occur during the conduct of the trial and result in noteworthy study protocol violations.



Sol-Gel Technologies Ltd. SGT-65-05


All efficacy analyses performed on the PP population will be according to the treatment they received.

# 8.5 Demographic and Other Baseline Characteristics

All Baseline summaries will be done on the ITT, PP, and Safety populations by treatment group and overall.

Sex, race, ethnicity, and Baseline IGA will be summarized by counts and percentages. Age, height (cm), weight (kg), body mass index (BMI), and Baseline lesion counts will be summarized with descriptive statistics.

Age, height, weight, BMI, and Baseline lesion counts will be compared among the two treatment groups using a two-way analysis of variance (ANOVA) with factors of treatment group and analysis center. Ethnicity, race, sex, and Baseline IGA will be analyzed with a Cochran-Mantel-Haenszel test stratified by analysis center.

Age will be calculated as the difference in days between the date of birth and the date of informed consent and converted to years by dividing the number of days by 365.25 and using a floor function to drop the decimal portion. In case the exact birth day is missing, day 15 will be used. The BMI will be calculated as weight (kg) divided by squared height (m<sup>2</sup>).

Medical histories will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary and presented in a by-subject listing.

The medical history data will be summarized with frequencies and percentages of patients with at least one medical history term reported, and patient frequencies and percentages on the System Organ Class (SOC) and Preferred Term (PT) levels. The number of events will also be summarized. The table will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of PT.

#### **8.6** Prior and Concomitant Medications

Concomitant medications will be coded to preferred name and Anatomical Therapeutic Chemical (ATC) classification of ingredients using the World Health Organization (WHO) Drug Global Dictionary, Format B3, Version March 1, 2018.

Medications which start prior to first application will be considered prior medications. Ongoing medications and medications ending after the date of first application will be considered concomitant medications. If the date of first application is unknown and the medication is not



Sol-Gel Technologies Ltd. SGT-65-05


listed as ongoing the interval will be considered "unknown". If the date of first application is unknown and the medication is listed as ongoing the interval will be considered concomitant.

Incomplete medication start and end dates will be imputed as described in Section 8.1.5.4

A summary of prior and concomitant medications will be provided.

A by-subject listing of all prior and concomitant medications will be presented for the Safety population.

## 8.7 Analysis of Efficacy

Inflammatory and non-inflammatory lesion counts will be summarized at each evaluation from Baseline through Week 12. Absolute and percent change in lesion counts will be summarized at Weeks 2, 4, 8, and 12. IGA scores will be summarized from Baseline through Week 12 using descriptive statistics. The dichotomized IGA scores will be summarized at Weeks 2, 4, 8, and 12 using descriptive statistics.

Primary, secondary, and supportive efficacy analyses will be conducted on the ITT (primary) population. Primary and secondary efficacy analyses will be conducted on the PP (supportive) population.

All efficacy results will be presented in by-subject listings.

# 8.7.1 Primary Efficacy Analysis

The primary efficacy analysis will be presented on both the ITT and PP populations.

## 8.7.1.1 Lesion Counts

Tests of superiority for the absolute change from Baseline in inflammatory and non-inflammatory lesions will be based on either parametric or non-parametric methods consistent with the statistical assumptions required to support the analyses. Specifically, the tests of superiority will be based on an ANCOVA with factors of treatment and analysis center and the respective Baseline lesion count as a covariate or on ranked data submitted to an ANCOVA with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. If the treatment-by-analysis center interaction effect is significant at an alpha less than 0.10, then the effect will be included in the model; otherwise it will be removed.

A skewness test, based on the methods presented by J.H. Zar [4], will be applied to the residuals resulting from an ANCOVA. A two-sided p-value for the skewness test significant at 0.01 will



Sol-Gel Technologies Ltd. SGT-65-05


imply the use of the non-parametric method. If a parametric analysis is indicated, the results of the parametric analysis will be considered the primary analysis. Should a non-parametric analysis be indicated, the absolute or percent changes in lesion counts will be rank transformed prior to submitting them to the ANCOVA. Results of the rank-transformed analyses then will be considered the primary analysis; however, results of the non-ranked transformed analyses will also be presented.

The following steps provide a brief synopsis of the process that will be followed.

- 1. Missing data will be imputed using multiple imputation. Refer to Section 8.1.5.1.
- 2. The pooling analysis will be conducted. Refer to Section 8.1.7.
  - a. The treatment-by-analysis center interaction p-values from both parametric and non-parametric (unranked and ranked) analyses will be presented, along with the skewness p-value calculated from the residuals from the unranked ANCOVA. The skewness p-value will determine which analysis results to report:
    - i. Skewness p-value > 0.01: Report results based on the parametric (unranked) approach.
    - ii. Skewness p-value  $\leq 0.01$ : Report results based on the non-parametric (ranked) approach.
- 3. For the primary efficacy analysis
  - a. Results of both parametric and non-parametric (unranked and ranked) analyses will be presented. For each, data will be submitted to an ANCOVA with factors of treatment and analysis center and Baseline lesion count as a covariate (if the treatment-by-analysis center interaction p-value is ≤ 0.10, the interaction will also be included in the model). The residuals from the unranked analysis will be used to calculate the skewness p-value. The skewness p-value will determine which analysis results to report:
    - i. Skewness p-value > 0.01: Report results from the parametric (unranked) ANCOVA.
    - ii. Skewness p-value  $\leq 0.01$ : Report results from the non-parametric (ranked) ANCOVA.
- 4. If there was a significant treatment by analysis center interaction (as determined in step 1 the pooling analysis), a sensitivity analysis will be performed as described in



Sol-Gel Technologies Ltd. SGT-65-05


Section 8.1.7 to find the extreme analysis center(s). Then step 3 above will be repeated the extreme analysis center(s) removed, to confirm the treatment response.

# 8.7.1.2 Investigator Global Assessment (IGA)

The IGA will be dichotomized into "success" and "failure" with a patient considered a success for those visits if the IGA is at least 2 grades less than Baseline and "Clear" or "Almost Clear". The analysis of the dichotomized IGA will be based on a logistic regression test with factors of treatment group and analysis center.

# 8.7.2 Sensitivity Efficacy Analysis

# 8.7.2.1 Sensitivity Analyses for Absolute Change in Lesion Count

## 8.7.2.1.1 Repeated Measures

The first sensitivity analyses for absolute change in lesion count (both inflammatory and non-inflammatory) will use a repeated measures ANCOVA, with treatment, analysis center, visit (i.e., Week 2, Week 4 and Week 8), and treatment group by visit interaction as independent factors and a covariate of Baseline lesion count. In this analysis, data from all post-baseline visits will be included with no imputation for missing data.

# **8.7.2.1.2 Model Based Multiple Imputation**

The second sensitivity analysis will use the model based multiple imputation method to impute missing data for the absolute change in lesion counts at Week 12. The multiple imputation will involve 3 principal tasks:

1. Missing values will be filled in 5 times to generate 5 complete data sets. The imputation model used will be an ANCOVA with factors of treatment group and analysis center, and a covariate of Baseline lesion count (i.e., the imputation model will be the same as the analysis model).

## Syntax:

```
proc mi data=datain out=dataout seed=&seed. nimpute=5 <options>;
  class trtpn sitegr1;
  var trtpn baseline sitegr1 week12;
  monotone logistic (sitegr1=trtpn baseline);
  monotone reg (week12=trtpn baseline sitegr1);
run;
```



Sol-Gel Technologies Ltd. SGT-65-05


2. Each complete data set will be analyzed with an ANCOVA with factors of treatment group, and analysis center, and a covariate of Baseline lesion count. Appropriate modifications will be made should the analysis be based on a non-parametric method.

3. Results from these analyses will be combined into a single inference.

Two random seeds will be needed to impute the inflammatory and non-inflammatory lesion counts. The following random seed has been pre-specified by using a random number generator:

Inflammatory Lesion Count Seed= 470857023

Non-inflammatory Lesion Count Seed= 2132132334

# **8.7.2.1.3 Tipping Point**

A tipping point analysis of the primary endpoints will be performed as a sensitivity analysis for the handling of missing data. The multiple imputation datasets used for the primary analyses will be used for the tipping point analyses for lesion counts. To perform the tipping point analysis, the imputed values from the multiple imputation datasets for only the E-BPO/E-ATRA cream arm will be adjusted, by adding a constant (shift value) to the lesion counts. Change from Baseline will then be recalculated with the changed imputed values. The shifted multiple imputed datasets will then be analyzed as described in the primary endpoint section. This will then be repeated by adding the constant again to create another new shifted multiple imputed dataset and that dataset will be analyzed. The resulting point estimates and p-values associated with each shift value will be presented in order to assess the magnitude of the shift value required to "tip" the p-value greater than 0.05.

# 8.7.2.2 Sensitivity Analyses for IGA

## 8.7.2.2.1 Repeated Measures

The first sensitivity analysis for the dichotomized IGA success will use a repeated measures logistic regression model (generalized estimating equations), with dichotomized IGA success as the dependent variable and treatment, analysis center, visit (i.e., Week 2, Week 4 and Week 8), and treatment group by visit interaction as independent factors. In this analysis, data from all post-baseline visits will be included with no imputation for missing data.



Sol-Gel Technologies Ltd. SGT-65-05


# **8.7.2.2.2 Model Based Multiple Imputation**

The second sensitivity analysis will use the model based multiple imputation method to impute missing data for the dichotomized IGA data. The multiple imputation will involve 3 principal tasks:

1. Missing values will be filled in 5 times to generate 5 complete data sets. The imputation model used logistic regression with factors of treatment group and analysis center (i.e., the imputation model will be the same as the analysis model).

Syntax:

```
proc mi data=datain out=dataout seed=&seed. nimpute=5 <options>;
  class trtpn sitegr1 diiga;
  var trtpn sitegr1 diiga;
  monotone logistic (sitegr1=trtpn);
  monotone logistic (diiga=trtpn sitegr1);
run;
```

- 2. Each complete data set will be analyzed with a logistic regression a factors of treatment group and analysis center.
- 3. Results from these analyses will be combined into a single inference.

One random seed will be needed to impute IGA. The following random seed has been prespecified by using a random number generator:

IGA Seed= 1497605671

# **8.7.2.2.3 Tipping Point**

A tipping point analysis of the primary endpoint will be performed as a sensitivity analysis for the handling of missing data. To perform the tipping point analysis for the dichotomized IGA, all combinations for the number of imputed successes for the nonrespondents in the E-BPO/E-ATRA cream group and the vehicle group will be analyzed to identify the points that would indicate a treatment failure using a p-value greater than 0.05. The resulting points of treatment failure will be plotted with the average number of successes in each treatment group from the primary multiple imputation analysis overlayed. The tipping points of the study will be identified by the points where the particular combinations of imputed successes that change the treatment success to a treatment failure.



Sol-Gel Technologies Ltd. SGT-65-05


# 8.7.3 Secondary Efficacy Analysis

Appropriate descriptive statistics will be computed for all secondary efficacy parameters.

Additionally, all inferential testing of percent change in lesions will follow the methods for the primary lesion count analyses. Methods corresponding to the analysis of IGA will be used to compare the proportion of patients in the E-BPO/EATRA Cream arm versus vehicle control achieving at least a 4-point reduction in pimples (item1 of the PRE-FACE) or in embarrassment (item5 of the PRE-FACE) scores from Baseline to Week 12.

A stepwise process will be conducted for testing the secondary efficacy endpoints in order to control for multiplicity, refer to Section 8.1.8.

The secondary efficacy analysis will be presented on the ITT and PP populations.

# 8.7.4 Supportive Efficacy Analysis

Appropriate descriptive statistics will be computed for all supportive efficacy parameters.

Additionally, all inferential testing will follow the methods for the co-primary variables wherein the continuous variables will parallel the lesion count analyses and the discrete dichotomized variables will follow the analysis of the IGA. Inferential testing for PGI-S and PGI-TS at Week 12 will use a cumulative logistic regression with factors of treatment group and analysis center. Missing values will not be imputed.

## 8.7.5 Exploratory Endpoint Analysis

The mean change in Acne-Qol domain scores from Baseline to Week 12 will be summarized using descriptive statistics.

Domain scores will be calculated as follows:

- 1. Code each response. Responses are numbered starting with 0 in ascending order.
  - For questions 1-14 and 18-19:
    - Extremely=0, Very Much=1, Quite A Bit=2, A Good Bit=3, Somewhat=4, A
       Little Bit=5, Not At All=6
  - For questions 15-17:
    - o 0=Extensive, 1=A Whole Lot, 2=A Lot, 3=A Moderate Amount, 4=Some, 5=Very Few, 6=None



Sol-Gel Technologies Ltd. SGT-65-05


- 2. Check for missing values and impute as follows:
  - Within each domain, a minimum number of responses is required in order to score the domain. At least 3 items must be answered within each domain in order to calculate the domain scores. If the minimum number of items have been answered but 1-2 questions have missing responses, calculate the mean value within the domain for the answered items and replace missing values with the mean value.
- 3. Calculate overall domain scores for each domain by summing the coded responses to each question in the domain.
  - Domains will be calculated as follows:
    - o Self-Perception domain calculated from questions 1, 2, 3, 6, and 10.
    - o Role-Emotional domain calculated from questions 4, 5, 7, 8, and 9.
    - o Role-Social domain calculated from questions 11, 12, 13, and 14.
    - o Acne Symptoms domain calculated from questions 15, 16, 17, 18, and 19.

# 8.8 Safety Evaluation

## 8.8.1 Extent of Exposure

The extent of exposure to study drug in each treatment group will be summarized by total number of days of exposure, total number of applications, number of missed applications and number and percentage of subjects who are compliant. A subject will be considered compliant with the dosing regimen if the subject applied 80% to 120% of the expected number of applications and did not miss more than 5 consecutive applications while enrolled in the study.

Days of exposure = Date of last study application – Date of first study application +1

The total number of applications taken is as follows:

(Date of Last Application – Date of First Application + 1) – (Number of Days marked as missed applications on the CRF) + (Number of extra applications marked on the CRF)

If a subject did apply medication on the last day, the total number of applications expected is as follows:

Date Subject End Participation – Date of Baseline +1.

If the total number of applications exceeds 89 then it will be set to 89.



Sol-Gel Technologies Ltd. SGT-65-05


If a subject did not apply medication on the last day, the total number of applications expected is as follows:

Date Subject End Participation - Date of Baseline

If the total number of applications exceeds 88 then it will be set to 88.

Compliance will be calculated as a percentage as 100 times the total number of applications taken from the first application until Week 12 divided by the total number of applications expected from first application until Week 12. Subjects who discontinue study medication before Week 12 will be considered to be 0% compliant for the number of days from discontinuing study medication until Week 12.

Compliance will not be calculated for subjects who are lost to follow-up or subjects who have unknown first or last application dates.

# 8.8.2 Adverse Events (AEs)

All AEs occurring during the study will be recorded and classified on the basis of MedDRA terminology. Descriptions of AEs will include the date of onset, the date the AE ended, the severity of the AE, the relationship to study product, the action taken regarding study product usage, the action taken to treat the AE, and the outcome. All reported TEAEs will be summarized by the number of patients reporting AEs, system organ class, severity, seriousness, and relationship to study product. TEAEs are those AEs with an onset on or after the date of the first study product application; if the AE is not indicated as prior to first application on the CRF then it will be considered a TEAE.

AEs will be summarized by treatment group and severity. Each patient will be counted only once within a system organ class or a preferred term by using the AEs with the highest severity within each category.

AEs will be summarized by treatment group and relationship to study product. Each patient will be counted only once within a system organ class or a preferred term by using the AEs with the greatest relationship within each category.

If relationship to study drug is reported as definitely, probably, or possible, then this is defined as related. If relationship to study drug is reported as unlikely or not related, then this is defined as unrelated.

Comparisons among treatment groups will be made by tabulating the frequency of patients with one or more AEs (classified into MedDRA terms) during the study. The Fisher's Exact test will


Sol-Gel Technologies Ltd. SGT-65-05


be used to compare the proportion of patients in each treatment group who report any AE at a significance level of 0.05. The specific system organ classes and preferred terms analyzed will be those that are reported by at least one percent of the patients in any treatment group.

All information pertaining to AEs noted during the study will be listed by patient, detailing verbatim given by the investigator, preferred term, system organ class, start date, stop date, severity, actions taken, and drug relatedness. The AE onset will also be shown relative (in number of days) to the day of initial application of the randomized study product.

Serious adverse events (SAEs) will be tabulated by patient within treatment groups.

In addition, a list of patients who discontinued from the study and a list of patients who experienced SAEs will also be provided.

### 8.8.1 Clinical Laboratory Evaluation

Urine pregnancy test results will be presented in a by-subject listing.

# 8.8.1 Other Observations Related to Safety

### **8.8.1.1** Cutaneous Safety Assessments

Descriptive statistics by treatment group and visit will be provided for pigmentation, erythema, dryness, and scaling.

### **8.8.1.2** Local Tolerability Assessments

Descriptive statistics by treatment group and visit will be provided for itching, burning and stinging.

## 8.8.1.3 Vital Signs

Vital sign measurements include heart rate (HR), sitting blood pressure (BP) (both systolic and diastolic), body temperature, and weight. The data will be summarized with descriptive statistics by visit and treatment group. In addition, the changes from baseline will be summarized with descriptive statistics.

Furthermore, to identify potentially clinically significant vital signs, the following criteria will be used and tabulated as a shift table by visit:

• Systolic Blood Pressure: <90 mmHg (low), 90-140 mmHg (normal), >140 mmHg (high)



Sol-Gel Technologies Ltd. SGT-65-05


• Diastolic Blood Pressure: <90 mm Hg (low), 90-100 mmHg (normal), >100 mmHg (high)

Heart Rate: <60 beats per minute (low), 60-100 beats per minute (normal), >100 beats per minute (high).

## 8.8.1.4 Physical Examination

Abnormal physical examination findings will be summarized by body system, visit, and treatment group. In addition to the summary, all physical examination findings will be listed.

#### 9. DETERMINATION OF SAMPLE SIZE

The following power calculations are based on the observed Week 12 results of the Phase 2 study, SGT-65-02. This study was a six-arm trial including S6G5T-3 and Vehicle Cream in the treatment of acne vulgaris. Estimates from the S6G5T-3 arm were used in the power assessments. The anticipated randomization ratio is 2:1 for S6G5T-3 and S6G5T-8 Vehicle Cream, respectively. The computations were performed with nQuery Advisor Version 7.0 using a two-sided test with a statistical significance value of 0.05.

A sample size of 274 in the S6G5T-3 and 137 in the Vehicle Cream group (total of 411) has 99% power to detect a statistically significant difference in inflammatory lesions. The estimated absolute change from Baseline in treatment means were -16.7 and -12.2 for S6G5T-3 and Vehicle Cream, respectively, with a common standard deviation of 10.0.

A sample size of 146 in the S6G5T-3 and 73 in the Vehicle Cream group (total of 219) has 99% power to detect a statistically significant difference in non-inflammatory lesions. The estimated absolute change from Baseline in treatment means were -23.7 and -13.7 for S6G5T-3 and Vehicle Cream, respectively, with a common standard deviation of 19.0.

A sample size of 231 in the S6G5T-3 and 116 in the Vehicle Cream has group (total of 346) has 99% power to detect a statistically significant difference the proportion of Patients who have at least a 2-grade reduction at Week 12 from Baseline in IGA and are Clear or Almost Clear. The estimated percentages with a 2-grade reduction at Week 12 from Baseline in the IGA and Clear or Almost Clear are 33.3% and 12.6% for S6G5T-3 and Vehicle Cream, respectively.

Therefore, a total of 420 Patients has adequate power to demonstrate statistical significance of S6GT5-3 over S6GT5-8 Vehicle Cream for the lesion count endpoints as well as dichotomized IGA.



Sol-Gel Technologies Ltd. SGT-65-05


#### 10. CHANGES IN THE PLANNED ANALYSES

There are no changes in the conduct of the study, but there are minor changes to the planned analyses.

Absolute change from Baseline in inflammatory and non-inflammatory lesion counts from Baseline to weeks 4 and 8 were removed from the supportive efficacy endpoints, as they were also included in the secondary efficacy endpoints.

The pooling analysis described in the protocol is updated in the statistical analysis plan (SAP) to reflect the intended analysis. The protocol discusses pooling sites with five or fewer subjects enrolled in each treatment arm. Taking into consideration the randomization ratio, the SAP requires ten subjects in the active treatment arm and five subjects in the vehicle group.

As part of the pooling analysis, the treatment effect within investigational site must be investigated. The protocol states the site main effect will be examined by using a one-way analysis of variance (for lesion count variables) or a logistic regression analysis (for dichotomized IGA) with a factor of site. The SAP instead explains site will be incorporated into the primary analysis models. Change from Baseline in lesion counts will be analyzed with an ANCOVA (unranked or ranked) with factors of treatment group, investigational site and treatment group by investigational site interaction, and the respective Baseline lesion count variable as a covariate. The dichotomized primary endpoint will be analyzed with a logistic regression with factors of treatment group, investigational site and the interaction term of treatment group by investigational site.

The protocol describes repeated measures sensitivity analyses for the primary efficacy endpoints. Treatment group, analysis center and visit are listed as factors for the repeated measures analyses. In addition to these factors, the SAP includes a factor of treatment group by visit interaction.

The protocol describes imputing only Week 12 data with MCMC imputation, but all missing post-Baseline data will be imputed.

The protocol provided did not provide seeds for the IGA MCMC imputation or for the model based multiple imputation, so those were added in the SAP. All seeds given the in SAP were produced in SAS as seeds given in the 65-05 protocol were identical to the 65-04 study protocol.

Geographic region was removed from the examination of subgroups as all sites in the study are in the United States.



Sol-Gel Technologies Ltd. SGT-65-05


An additional age grouping of 9-11 years, 12-17 years, 18-30 years, and 31 years and older was added to the subgroup summaries.

The secondary efficacy analysis wil be presented on the PP population in addition to the ITT population as specified in the protocol.

#### 11. REFERENCES

- 1. Bhate K, Williams HC. Epidemiology of acne vulgaris. Br J Dermatol. 2013Mar;168(3):474-485.
- 2. Gollnick H, Cunliffe W Berson D, et al; Global Alliance to Improve Outcomes in Acne. Management of acne: a report form a Global Alliance to Improve Outcomes in Acne. J Am Acad Dermatol. 2003;49(suppl 1):S1-S37.
- 3. Leyden J, Kaidbey K, Levy SF. The combination formulation of clindamycin 1% plus benzoyl peroxide 5% versus 3 different formulations of topical clindamycin alone in the reduction of Propionibacterium acnes. Am J Clin Dermatol 2001;2 (4):63-266.
- 4. Zar, JH. Bio-statistical analysis, 1984 2nd ed. Englewood Cliffs (NJ)Prentice-Hall.



**Statistical Analysis Plan** Sol-Gel Technologies Ltd. SGT-65-05

Version: 2

Date: 26 NOV 2019

# 12. INDEX OF PLANNED TABLES

| Table 14.0.1: Summary of Subject Completion/Discontinuation (All Randomized Subjects)44 |
|---|
| Table 14.0.2.1: Summary of Subject Enrollment and Evaluability (All Randomized Subjects)45 |
| Table 14.0.2.2: Summary of Subject Evaluability by Analysis Center and Investigational Site (All Randomized Subjects) |
| Table 14.1.1.1: Summary of Subject Demographic Characteristics (Intent-to-<br>Treat Population) |
| Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population)49 |
| Table 14.1.1.3: Summary of Subject Demographics (Safety Population)49 |
| Table 14.1.2.1: Subject Baseline Characteristics (Intent-to-Treat Population)50 |
| Table 14.1.2.2: Subject Baseline Characteristics (Per-Protocol Population)51 |
| Table 14.1.2.3: Subject Baseline Characteristics (Safety Population)51 |
| Table 14.1.3.1: Summary of Medical History by System Organ Class and Preferred Term (Intent-to-Treat Population) |
| Table 14.1.3.2: Summary of Medical History by System Organ Class and Preferred Term (Per-Protocol Population) |
| Table 14.1.3.3: Summary of Medical History by System Organ Class and Preferred Term (Safety Population) |
| Table 14.1.4.1: Summary of Prior Medications by ATC Level 2 and Preferred Name (Safety Population) |
| Table 14.1.4.2: Summary of Concomitant Medications by ATC Level 2 and Preferred Name (Safety Population) |
| Table 14.2.1.1: Pooling Analysis for Primacy Efficacy Endpoints (Intent-to-Treat Population)55 |
| Table 14.2.1.2: Primary Efficacy Analysis: Absolute Change from Baseline in Lesion Counts and Dichotomized IGA Success at Week 12 (Intent-to-Treat Population) |
| Table 14.2.1.3: Primary Efficacy Analysis: Absolute Change from Baseline in Lesion Counts and Dichotomized IGA Success at Week 12 (Per-Protocol Population) |
| Table 14.2.2.1.1: Summary of Inflammatory Lesion Counts at Each Evaluation (Intent-to-<br>Treat Population) |
| Table 14.2.2.1.2: Summary of Inflammatory Lesion Counts at Each Evaluation (Per-Protocol Population) |



**Statistical Analysis Plan** Sol-Gel Technologies Ltd. SGT-65-05

Version: 2

Date: 26 NOV 2019

| Table 14.2.2.2: Summary of Absolute Change in Inflammatory Lesion Counts at Week 12 by Analysis Center (Intent-to-Treat Population) |
|---|
| Table 14.2.3.1.1: Summary of Non-Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population) |
| Table 14.2.3.1.2: Summary of Non-Inflammatory Lesion Counts at Each Evaluation (Per-Protocol Population) |
| Table 14.2.3.2: Summary of Absolute Change in Non-Inflammatory Lesion Counts at Week 12 by Analysis Center (Intent-to-Treat Population)69 |
| Table 14.2.4.1.1: Summary of Investigator Global Assessment at Each Evaluation (Intent-to-Treat Population) |
| Table 14.2.4.1.2: Summary of Investigator Global Assessment at Each Evaluation (Per-Protocol Population) |
| Table 14.2.4.2: Summary of Investigator Global Assessment (Two Grade Reduction from Baseline and Clear or Almost Clear) at Week 12 by Analysis Center (Intent-to-Treat Population) |
| Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population)76 |
| Table 14.2.6.1: Sensitivity Analysis of Primary Endpoints: Absolute Change from Baseline in Lesion Counts and Dichotomized IGA Success at Week 12 (Intent-to- Treat Population) |
| Table 14.2.7.1: Sensitivity Tipping-Point Analysis of the Primary Endpoint: Lesion Counts at Week 12 (Intent-to-Treat Population) |
| Table 14.2.8.1: Secondary Efficacy Analyses (Intent-to-Treat Population) |
| Table 14.2.8.2: Secondary Efficacy Analyses (Per-Protocol Population) |
| Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)90 |
| Table 14.2.9.2: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Per-Protocol Population) |
| Table 14.2.10.1: Supportive Efficacy Analyses: PGI-TS, PGI-S, and PGI-C at Week 12 (Intent-to-Treat Population) |
| Table 14.2.11.1: Supportive Efficacy Analyses: Lesion Count and IGA119 |
| Table 14.2.12.1: Supportive Efficacy Analyses: PRE-FACE ASD Scores |
| Table 14.2.13.1: Supportive Efficacy Analyses: PRE-FACE AID Scores |
| Table 14.2.14.1: Summary of Patient Global Impression of Change (PGI-C) at Each Evaluation (Intent-to-Treat Population) |



**Statistical Analysis Plan** Sol-Gel Technologies Ltd. SGT-65-05

Version: 2

Date: 26 NOV 2019

| Table 14.2.15.1: Summary of Patient Global Impression of Symptom Severity (PGI-S) at Eac<br>Evaluation (Intent-to-Treat Population) | |
|---|---|
| Table 14.2.16.1: Summary of Patient Global Impression of Treatments Satisfaction (PGI-TS) Each Evaluation (Intent-to-Treat Population) | |
| Table 14.2.17.1: Summary of Acne-QoL Questionnaire Responses at Baseline and Week 12 (Intent-to-Treat Population) | 134 |
| Table 14.3.0.1: Summary of Extent of Exposure (Safety Population) | 138 |
| Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population) | 139 |
| Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) | 153 |
| Table 14.3.1.2.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Or Class and Preferred Term (Safety Population) | |
| Table 14.3.1.2.3: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population) | 156 |
| Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug (Safety Population) | |
| Table 14.3.1.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) | 158 |
| Table 14.3.1.3.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) | 160 |
| Table 14.3.1.3.3: Summary of Serious Treatment-Emergent Adverse Events by Severity (Safety Population) | 161 |
| Table 14.3.1.3.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship Study Drug (Safety Population) | |
| Table 14.3.1.4: Summary of Vital Signs (Safety Population) | 163 |
| Table 14.3.1.4.2: Shift Table of Vital Signs (Safety Population) | 168 |
| Table 14.3.1.5: Summary of Abnormal Physical Examination Findings by Visit (Safety Population) | 169 |
| Table 14.3.1.6: Summary of Patient Global Impression of Treatment Side-Effects (PGI-SE) a Each Evaluation (Safety Population) | |



Table 14.0.1: Summary of Subject Completion/Discontinuation (All Randomized Subjects)

| | E-BPO/E-ATRA 3%/0.1% Cream | Vehicle Cream | Total |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Completed Study | | | |
| Yes | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Reason for Discontinuation | | | |
| Adverse Event | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost to Follow-Up | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lack of Efficacy | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pregnancy | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Protocol Violation | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Withdrawal by Parent/Guardian | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Withdrawal by Subject | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Study Terminated by Sponsor | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Physician Decision | xx = (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Worsening of Condition | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx = (xx.x%) | xx (xx.x%) | xx ( xx.x%) |



Table 14.0.2.1: Summary of Subject Enrollment and Evaluability (All Randomized Subjects)

| | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Number of Randomized Subjects | XX | XX | XX |
| Number of Subjects Included in the ITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the ITT Population Reason Excluded from the ITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Dispensed Study Drug | XX (XX.X%) | XX (XX.X%) | xx ( xx.x%) |
| Number of Subjects Included in the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the Safety Population<br>Reasons Excluded from the Safety Population <sup>a</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Documented use of Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No Post-Baseline Safety Assessment | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| Number of Subjects Included in the PP Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Subjects Excluded from the PP Population Reasons Excluded from the PP Population <sup>a</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Included in ITT Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Violated Inclusion/Exclusion Criteria | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Used Interfering Concomitant Medication | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Did not Attend Week 12/ET Visit | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missed More Than 1 Post-Baseline Visit Prior to Week 12 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Compliant with Dosing Regimen <sup>b</sup> | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Week 12/ET Visit Out of Window (+/-4 days) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Table includes primary reason (assigned in order presented in table) for reason subject was excluded.

b Subjects lost to follow-up not included. A subject was considered compliant with the dosing regimen if the subject applied 80-120% of the expected number of applications and did not miss more than 5 consecutive applications while enrolled in the study.



Table 14.0.2.2: Summary of Subject Evaluability by Analysis Center and Investigational Site
(All Randomized Subjects)

| | | E-BPO/E-ATRA 3%/0.1% Cream | | Vehicle Cream | | | | |
|---|---|---|---|---|---|---|---|---|
| Analysis<br>Center | Investigational Site | Number<br>Randomized | ITT | PP | Safety | ITT | PP | Safety |
| XX | XX | XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | XX | XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | XX | XX | XX | XX | XX | XX | XX | XX |
| | XX | XX | XX | XX | XX | XX | XX | XX |



Table 14.1.1.1: Summary of Subject Demographic Characteristics (Intent-to-Treat Population) 

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Total<br>(N=xxx) | P-Value |
|---|---|---|---|---|
| Age (years) | | | | |
| n | XX | XX | XX | x.xxx <sup>a</sup> |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | |
| < Median (xx years) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | |
| ≥ Median (xx years) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | |
| < 18 years | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | |
| ≥ 18 years and < Median (xx years) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| ≥ Median (xx years) | XX (XX.X%) | xx (xx.x%) | xx ( xx.x%) | |
| 9-11 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| 12-17 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| 18-30 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| ≥ 31 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |

P-value from a two-way analysis of variance with factors of treatment group and analysis center.
 P-value from a Cochran-Mantel-Haenszel general association test, stratified by analysis center.

<sup>&</sup>lt;sup>c</sup> See Listing 16.2.4.1 for a complete list of other races.



Table 14.1.1.1: Summary of Subject Demographics (Intent-to-Treat Population) 

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Total<br>(N=xxx) | P-Value |
|---|---|---|---|---|
| Sex | | | | L. |
| n | XX | XX | XX | $x.xxx^b$ |
| Male | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | |
| Female | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | | | | |
| n | XX | XX | XX | $x.xxx^b$ |
| Hispanic or Latino | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | |
| Race | | | | |
| n | XX | XX | xx | $x.xxx^b$ |
| American Indian or Alaska Native | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| Asian | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| Multiple/Other <sup>c</sup> | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |

Repeat Table 14.1.1.1 for the following tables:

P-value from a two-way analysis of variance with factors of treatment group and analysis center.
 P-value from a Cochran-Mantel-Haenszel general association test, stratified by analysis center.
 See Listing 16.2.4.1 for a complete list of other races.



Table 14.1.1.2: Summary of Subject Demographics (Per-Protocol Population)
Table 14.1.1.3: Summary of Subject Demographics (Safety Population)



Table 14.1.2.1: Subject Baseline Characteristics (Intent-to-Treat Population) 

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Total<br>(N=xxx) | P-Value |
|---|---|---|---|---|
| Height (cm) | | | | |
| n | XX | XX | XX | x.xxx <sup>a</sup> |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | |
| Weight (kg) | | | | |
| n | XX | XX | XX | x.xxx <sup>a</sup> |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | |
| BMI (kg/m²) | | | | |
| n | XX | XX | XX | x.xxx <sup>a</sup> |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | |

P-value from a two-way analysis of variance with factors of treatment group and analysis center.
 P-value from a Cochran-Mantel-Haenszel general association test, stratified by analysis center.



Table 14.1.2.1: Subject Baseline Characteristics (Intent-to-Treat Population) 

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Total<br>(N=xxx) | P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count | | | | |
| n | XX | XX | XX | $\mathbf{X.XXX}^{\mathbf{a}}$ |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | |
| Non-Inflammatory Lesion Count | | | | |
| n | XX | XX | XX | $\mathbf{X.XXX}^{\mathbf{a}}$ |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.XX | XX.XX | XX.XX | |
| Median | XX.X | XX.X | XX.X | |
| Min. to Max. | xx to xx | xx to xx | xx to xx | |
| Investigator Global Assessment | | | | |
| n | XX | XX | XX | $x.xxx^b$ |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| 1 – Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | |

Repeat Table 14.1.2.1 for the following table:

Table 14.1.2.2: Subject Baseline Characteristics (Per-Protocol Population)

Table 14.1.2.3: Subject Baseline Characteristics (Safety Population)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

P-value from a two-way analysis of variance with factors of treatment group and analysis center.
 P-value from a Cochran-Mantel-Haenszel general association test, stratified by analysis center.



Table 14.1.3.1: Summary of Medical History by System Organ Class and Preferred Term (Intent-to-Treat Population)

| System Organ Class Preferred Term | E-BPO/E-<br>3%/0.1%<br>(N=x: | Cream | | e Cream<br>=xxx) | | otal<br>xxx) |
|---|---|---|---|---|---|---|
| Number (%) of Subjects Reporting at Least One Medical History Term | | By Event <sup>b</sup> | By Subject <sup>a</sup><br>xx (xx.x%) | By Event <sup>b</sup> | By Subject <sup>a</sup><br>xx (xx.x%) | By Event <sup>b</sup> |
| System Organ Class<br>Preferred Term | xx (xx.x%)<br>xx (xx.x%) | | xx ( xx.x%)<br>xx ( xx.x%) | | xx ( xx.x%)<br>xx ( xx.x%) | |

Note: MedDRA Version 21.0

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

{NOTE TO PROGRAMMER: The table will be sorted by overall descending frequency of SOC and then, within a SOC, by overall descending frequency of PT}

Repeat Table 14.1.3.1 for the following table:

Table 14.1.3.2: Summary of Medical History by System Organ Class and Preferred Term (Per-Protocol Population)

Table 14.1.3.3: Summary of Medical History by System Organ Class and Preferred Term (Safety Population)

<sup>&</sup>lt;sup>a</sup> Counts reflect number of subjects reporting one or more medical history terms that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once. Percentages are based on the number of subjects in the safety population.

<sup>&</sup>lt;sup>b</sup> Counts reflect number of medical history terms that map to MedDRA.



Table 14.1.4.1: Summary of Prior Medications by ATC Level 2 and Preferred Name (Safety Population)

| ATC Level 2 Term <sup>a</sup> Preferred Name | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Number (%) of Subjects Reporting at Least One Prior Medication | xx ( xx.x%) | xx ( xx.x%) |
| ATC Level 2 Term Preferred Name | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |

Note: WHO Drug Global Dictionary, Format B3, Version March 1, 2018
Prior medications are those used before the date of first study drug application.

<sup>&</sup>lt;sup>a</sup> Counts reflect number of subjects reporting one or more medications that map to the WHO term. At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once. Percentages are based on the number of subjects in the safety population.



Table 14.1.4.2: Summary of Concomitant Medications by ATC Level 2 and Preferred Name (Safety Population)


| ATC Level 2 Term <sup>a</sup> Preferred Name | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Number (%) of Subjects Reporting at Least One Concomitant Medication | xx ( xx.x%) | xx ( xx.x%) |
| ATC Level 2 Term Preferred Name | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |

Note: WHO Drug Global Dictionary, Format B3, Version March 1, 2018

Concomitant medications are those used on/after the date of first study drug application.

<sup>&</sup>lt;sup>a</sup> Counts reflect number of subjects reporting one or more medications that map to the WHO term. At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once. Percentages are based on the number of subjects in the safety population.



Table 14.2.1.1: Pooling Analysis for Primacy Efficacy Endpoints (Intent-to-Treat Population)

| | Investigational S | Site Pooling Analysis Investigational | Analysis Cent | er Pooling Analysis Analysis Center |
|---|---|---|---|---|
| | Skewness | Site by Treatment | Skewness | Treatment |
| Endpoint Absolute Change from Baseline in Inflammatory Lesion Counts at Week 12 | P-Value<br>x.xxx <sup>c</sup> | Group P-Value | P-Value<br>x.xxx <sup>c</sup> | Group P-Value |
| Ranked Analysis | | X.XXX <sup>a</sup> | | x.xxx <sup>e</sup> |
| Unranked Analysis | | $x.xxx^b$ | | $\mathbf{x}.\mathbf{x}\mathbf{x}^{\mathbf{f}}$ |
| Absolute Change from Baseline in Non-Inflammatory Lesion Counts at Week 12 | x.xxx <sup>c</sup> | | x.xxx <sup>c</sup> | |
| Ranked Analysis | | X.XXX <sup>a</sup> | | x.xxx <sup>e</sup> |
| Unranked Analysis | | X.XXX <sup>b</sup> | | $\mathbf{X}.\mathbf{X}\mathbf{X}\mathbf{X}^{\mathrm{f}}$ |
| Two Grade Reduction from Baseline in IGA and Achieving Clear or Almost Clear at Week 12 | NA | x.xxx <sup>d</sup> | NA | x.xxx <sup>g</sup> |

<sup>&</sup>lt;sup>a</sup> P-value for the interaction term from a ranked analysis of covariance with factors of treatment, investigational site, treatment by investigational site interaction and the respective Baseline lesion count as a covariate.

Note: Multiple imputation (MCMC) used to impute missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

{NOTE TO PROGRAMMER: ADJUST FOOTNOTE "d" AND/OR "g" IF FIRTH'S PENALIZED LIKELIHOOD IS NEEDED}

<sup>&</sup>lt;sup>b</sup> P-value for the interaction term from an unranked analysis of covariance with factors of treatment, investigational site, treatment by investigational site interaction and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>c</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset. The average p-value is presented.

<sup>&</sup>lt;sup>d</sup> P-value for the interaction term from a logistic regression with factors of treatment, investigational site, treatment by investigational site interaction.

<sup>&</sup>lt;sup>e</sup> P-value for the interaction term from a ranked analysis of covariance with factors of treatment, analysis center, treatment by analysis center interaction and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>f</sup> P-value for the interaction term from an unranked analysis of covariance with factors of treatment, analysis center, treatment by analysis center interaction and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>g</sup> P-value for the interaction term from a logistic regression with factors of treatment, analysis center, treatment by analysis center interaction.



Table 14.2.1.2: Primary Efficacy Analysis: Absolute Change from Baseline in Lesion Counts and Dichotomized IGA Success at Week 12 (Intent-to-Treat Population)

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Skewness<br>P-Value | Treatment P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count – Absolute Change | | | | |
| from Baseline | | | _ | |
| LSMean <sup>a</sup> | XX.X | XX.X | x.xxx <sup>b</sup> | X.XXX <sup>a</sup> |
| $LSSD^a$ | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| Non-Inflammatory Lesion Count – Absolute Chang from Baseline | е | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| LSSD <sup>a</sup> | XX.XX | XX.XX | | X.XXX <sup>c</sup> |
| At Least Two Grade Reduction from Baseline and<br>Achieving Clear or Almost Clear | | | | |
| Success | xx.x% | xx.x% | N/A | $\mathbf{x}.\mathbf{x}\mathbf{x}\mathbf{x}^{\mathbf{d}}$ |
| Failure | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> | | |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (MCMC) used to impute missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

{NOTE TO PROGRAMMER: ADJUST FOOTNOTE "d" IF FIRTH'S PENALIZED LIKELIHOOD IS NEEDED}

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset. The average p-value is presented.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Repeat Table 14.2.1.2 for the following table:

Table 14.2.1.3: Primary Efficacy Analysis: Absolute Change from Baseline in Lesion Counts and Dichotomized IGA Success at Week 12 (Per-Protocol Population)

Update footnote to "Note: Missing values imputed using last observation carried forward."



Table 14.2.2.1.1: Summary of Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population)


| Inflammatory Lesion Counts | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.2.2.1.1: Summary of Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population)


| Inflammatory Lesion Counts Week 4 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.2.2.1.1: Summary of Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population)


| <b>Inflammatory Lesion Counts</b> Week 8 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.2.2.1.1: Summary of Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population)


| Inflammatory Lesion Counts Week 12 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics for Weeks 2, 4, 8, and 12 represent average values, obtained from averaging the summary statistics generated from each imputed dataset. Negative values represent decrease from Baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Table 14.2.2.1.1 for the following table:

Table 14.2.2.1.2: Summary of Inflammatory Lesion Counts at Each Evaluation (Per-Protocol Population)

Change footnote to "Note: Missing values imputed using last observation carried forward. Negative values represent decrease from Baseline."



Table 14.2.2.2: Summary of Absolute Change in Inflammatory Lesion Counts at Week 12 by Analysis Center (Intent-to-Treat Population)

| | E-BPO/E- | ATRA 3%/0.1<br>(N=xxx) | % Cream | , | Vehicle Cream (N=xxx) | |
|---|---|---|---|---|---|---|
| Analysis Center (Investigational Sites) | <u>n</u> | Mean | SD | n | Mean | SD |
| xx(y, z) | XX | XX.X | XX.XX | XX | XX.X | XX.XX |
| xx(y, z) | XX | XX.X | XX.XX | XX | XX.X | XX.XX |
| xx(y, z) | XX | XX.X | XX.XX | XX | XX.X | XX.XX |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained from averaging the summary statistics generated from each imputed dataset. Negative values represent decrease from Baseline.



Table 14.2.3.1.1: Summary of Non-Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population)


| Non-Inflammatory Lesion Counts | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.2.3.1.1: Summary of Non-Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population) 

| Non-Inflammatory Lesion Counts<br>Week 4 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| | XX | XX |
| n<br>Mean | | |
| SD | XX.X | XX.X |
| | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.2.3.1.1: Summary of Non-Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population)


| Non-Inflammatory Lesion Counts<br>Week 8 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.2.3.1.1: Summary of Non-Inflammatory Lesion Counts at Each Evaluation (Intent-to-Treat Population)


| Non-Inflammatory Lesion Counts | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Percent Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics for Weeks 2, 4, 8, and 12 represent average values, obtained from averaging the summary statistics generated from each imputed dataset. Negative values represent decrease from Baseline.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Repeat Table 14.2.3.1.1 for the following table:

Table 14.2.3.1.2: Summary of Non-Inflammatory Lesion Counts at Each Evaluation (Per-Protocol Population)

Change footnote to "Note: Missing values imputed using last observation carried forward. Negative values represent decrease from Baseline."



Table 14.2.3.2: Summary of Absolute Change in Non-Inflammatory Lesion Counts at Week 12 by Analysis Center (Intent-to-Treat Population)

| | E-BPO/E- | ATRA 3%/0.1<br>(N=xxx) | % Cream | , | Vehicle Cream (N=xxx) | |
|---|---|---|---|---|---|---|
| Analysis Center (Investigational Sites) | <u>n</u> | Mean | SD | n | Mean | SD |
| xx(y, z) | XX | XX.X | XX.XX | XX | XX.X | XX.XX |
| xx(y, z) | XX | XX.X | XX.XX | XX | XX.X | XX.XX |
| xx(y, z) | XX | XX.X | XX.XX | XX | XX.X | XX.XX |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained from averaging the summary statistics generated from each imputed dataset. Negative values represent decrease from Baseline.



Table 14.2.4.1.1: Summary of Investigator Global Assessment at Each Evaluation (Intent-to-Treat Population)


| Investigator Global Assessment | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| 0 - Clear | XX.X% | xx.x% |
| 1 - Almost Clear | XX.X% | xx.x% |
| 2 - Mild | XX.X% | xx.x% |
| 3 - Moderate | XX.X% | xx.x% |
| 4 - Severe | xx.x% | XX.X% |



Table 14.2.4.1.1: Summary of Investigator Global Assessment at Each Evaluation (Intent-to-Treat Population)


| Investigator Global Assessment | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 4 | 0/ | 0/ |
| 0 - Clear | XX.X% | XX.X% |
| 1 - Almost Clear | XX.X% | xx.x% |
| 2 - Mild | XX.X% | XX.X% |
| 3 - Moderate | XX.X% | XX.X% |
| 4 - Severe | XX.X% | XX.X% |
| Two Grade Reduction from Baseline | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | $XX.X^{0}/_{0}$ |
| Failure | xx.x% | XX.X% |
| Two Grade Reduction from Baseline and Achieving Clear or Almost Clear | | |
| Success | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% |



Table 14.2.4.1.1: Summary of Investigator Global Assessment at Each Evaluation (Intent-to-Treat Population)


| Investigator Global Assessment | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 8 | | |
| 0 - Clear | xx.x% | xx.x% |
| 1 - Almost Clear | xx.x% | xx.x% |
| 2 - Mild | xx.x% | xx.x% |
| 3 - Moderate | xx.x% | xx.x% |
| 4 - Severe | xx.x% | xx.x% |
| Two Grade Reduction from Baseline | | |
| Success | xx.x% | xx.x% |
| Failure | xx.x% | XX.X% |
| Two Grade Reduction from Baseline and Achieving Clear or Almost Clear | | |
| Success | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% |


Table 14.2.4.1.1: Summary of Investigator Global Assessment at Each Evaluation (Intent-to-Treat Population)


| Investigator Global Assessment | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 12<br>0 - Clear | xx.x% | xx.x% |
| 1 - Almost Clear | | |
| | XX.X% | xx.x% |
| 2 - Mild | xx.x% | xx.x% |
| 3 - Moderate | XX.X% | $XX.X^{0/0}$ |
| 4 - Severe | xx.x% | xx.x% |
| Two Grade Reduction from Baseline | | |
| Success | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% |
| Two Grade Reduction from Baseline and Achieving Clear or Almost Clear | | |
| Success | xx.x% | $xx.x^{0}/_{0}$ |
| Failure | xx.x% | xx.x% |

Note: Multiple imputation (MCMC) used to impute missing values. Percentages for Weeks 2, 4, 8, and 12 represent average values, obtained from averaging the summary statistics generated from each imputed dataset.



Repeat Table 14.2.4.1.1 for the following table:

Table 14.2.4.1.2: Summary of Investigator Global Assessment at Each Evaluation (Per-Protocol Population)

Change footnote to "Note: Missing values imputed using last observation carried forward."



Table 14.2.4.2: Summary of Investigator Global Assessment (Two Grade Reduction from Baseline and Clear or Almost Clear) at Week 12 by Analysis Center (Intent-to-Treat Population)

| | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Analysis Center (Investigational Sites) | XX.X% | XX.X% |
| xx(y,z) | xx.x% | xx.x% |
| xx(y,z) | xx.x% | xx.x% |
| xx(y, z) | xx.x% | xx.x% |
| xx(y, z) | xx.x% | XX.X% |
| xx(y, z) | XX.X% | XX.X% |
| xx(y, z) | XX.X% | XX.X% |
| xx(y, z) | xx.x% | XX.X% |
| xx(y, z) | XX.X% | xx.x% |
| xx(y, z) | xx.x% | xx.x% |

Note: Multiple imputation (MCMC) used to impute missing values. Summary statistics represent average values, obtained from averaging the summary statistics generated from each imputed dataset.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Age | $_{\text{def}} < \text{Median Age } (xx)$ | | Age >= Median Age (xx) | |
|---|---|---|---|---|
| 9 | E-BPO/E-ATRA | | E-BPO/E-ATRA | • , , |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | (N=xxx) | N=xxx | (N=xxx) | N=xxx |
| Inflammatory Lesion Count – Absolute Change from Baseline | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Chang from Baseline | ge | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Two Grade Reduction from Baseline in IGA and<br>Achieving Clear or Almost Clear | | | | |
| | XX.X% | XX.X% | XX.X% | XX.X <sup>0</sup> / <sub>0</sub> |
| Success | ΛΛ.Λ/0 | 7171.7170 | | |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Age | Age | < 18 | $\phantom{aaaaaaaaaaaaaaaaaaaaaaaaaaaaaaaaaaa$ | |
|---|---|---|---|---|
| | E-BPO/E-ATRA | | E-BPO/E-ATRA | • , |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | N=xxx | (N=xxx) | N=xxx | N=xxx |
| Inflammatory Lesion Count – Absolute Change | | | | |
| from Baseline | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Chan | re. | | | |
| from Baseline | ge | | | |
| n | xxx | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | | | | |
| SD<br>Median | | | xx x | |
| Median | XX.X | XX.X | XX.X<br>xx to xx | XX.X |
| | | | xx.x<br>xx to xx | |
| Median | XX.X | XX.X | | XX.X |
| Median Min. to Max. Two Grade Reduction from Baseline in IGA and | XX.X | XX.X | | XX.X |
| Median<br>Min. to Max. | XX.X | XX.X | | XX.X |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Age | 9-11 | years | 12-17 | years |
|---|---|---|---|---|
| | E-BPO/E-ATRA | , | E-BPO/E-ATRA | • |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | (N=xxx) | (N=xxx) | (N=xxx) | N=xxx |
| Inflammatory Lesion Count – Absolute Change from Baseline | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Chan from Baseline | ge | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Two Grade Reduction from Baseline in IGA and | | | | |
| Achieving Clear or Almost Clear | | | | |
| Achieving Clear or Almost Clear<br>Success | XX.X% | xx.x% | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Age | 18-30 | years | >= 31 | years |
|---|---|---|---|---|
| | E-BPO/E-ATRA | • | E-BPO/E-ATRA | • |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | (N=xxx) | (N=xxx) | (N=xxx) | N=xxx |
| Inflammatory Lesion Count – Absolute Change from Baseline | | | · | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Change from Baseline | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Two Grade Reduction from Baseline in IGA and | | | | |
| Achieving Clear or Almost Clear<br>Success | $XX.X^{0}/_{0}$ | XX.X% | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> |
| Failure | xx.x% | xx.x% | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Sex | Male | | Female | |
|---|---|---|---|---|
| | E-BPO/E-ATRA | | E-BPO/E-ATRA | |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | N=xxx | (N=xxx) | (N=xxx) | (N=xxx) |
| Inflammatory Lesion Count – Absolute Change from Baseline | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Chan from Baseline | ge | | | |
| n | xxx | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Two Grade Reduction from Baseline in IGA and | | | | |
| Achieving Clear or Almost Clear | | | | |
| Success | XX.X% | XX.X% | XX.X% | xx.x% |
| Failure | XX.X% | XX.X% | XX.X% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Ethnicity <sup>a</sup> | Hispanic | or Latino | Not Hispanic or Latino | |
|---|---|---|---|---|
| • | E-BPO/E-ATRA | | E-BPO/E-ATRA | |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | (N=xxx) | (N=xxx) | N=xxx | (N=xxx) |
| Inflammatory Lesion Count – Absolute Change from Baseline | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | xx.xx | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Change from Baseline | | | | |
| n | XXX | XXX | xxx | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Two Grade Reduction from Baseline in IGA and | | | | |
| Achieving Clear or Almost Clear | 0.4 | 0./ | 0.4 | 0.1 |
| Success | XX.X% | XX.X% | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Race | Wh | ite | Non-V | White |
|---|---|---|---|---|
| | E-BPO/E-ATRA | | E-BPO/E-ATRA | |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | (N=xxx) | (N=xxx) | N=xxx | (N=xxx) |
| Inflammatory Lesion Count – Absolute Change | | | | |
| from Baseline | | | | |
| n | xxx | XXX | xxx | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Chan | σe | | | |
| from Baseline | 50 | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Two Grade Reduction from Baseline in IGA and | | | | |
| Two Grade Reduction from Baseline in IGA and Achieving Clear or Almost Clear | | | | |
| Two Grade Reduction from Baseline in IGA and<br>Achieving Clear or Almost Clear<br>Success | xx.x% | xx.x% | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.5.1: Subgroup Summaries of Primary Endpoints (Intent-to-Treat Population) 

| Baseline IGA | Mode | erate | Sev | ere |
|---|---|---|---|---|
| | E-BPO/E-ATRA | | E-BPO/E-ATRA | |
| | 3%/0.1% Cream | Vehicle Cream | 3%/0.1% Cream | Vehicle Cream |
| | N=xxx | N=xxx | N=xxx | (N=xxx) |
| Inflammatory Lesion Count – Absolute Change | | | · | |
| from Baseline | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Non-Inflammatory Lesion Count – Absolute Cl<br>from Baseline | nange | | | |
| n | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Two Grade Reduction from Baseline in IGA an Achieving Clear or Almost Clear | d | | | |
| Two Grade Reduction from Baseline in IGA an<br>Achieving Clear or Almost Clear<br>Success | d<br>xx.x% | xx.x% | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Ethnicities of Not Reported and Unknown are not included.



Table 14.2.6.1: Sensitivity Analysis of Primary Endpoints: Absolute Change from Baseline in Lesion Counts and Dichotomized IGA Success at Week 12

(Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Skewness<br>P-Value | Treatment P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count – Absolute Change | | | | |
| from Baseline | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| LSSD <sup>a</sup> | xx.xx | XX.XX | | x.xxx <sup>c</sup> |
| Non-Inflammatory Lesion Count – Absolute Change<br>from Baseline<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| At Least Two Grade Reduction from Baseline and<br>Achieving Clear or Almost Clear<br>Success<br>Failure | xx.x%<br>xx.x% | xx.x%<br>xx.x% | N/A | x.xxx <sup>d</sup> |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from a repeated measures analysis of covariance with factors of treatment group, analysis center, visit and treatment group by visit interaction, and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

<sup>&</sup>lt;sup>b</sup> Skewness test based on methods presented by J.H. Zar (1984).

<sup>&</sup>lt;sup>c</sup> P-value from a ranked repeated measures analysis of covariance with factors of treatment group, analysis center, visit and treatment group by visit interaction, and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a repeated measures logistic regression with factors of treatment group, analysis center, visit and treatment group by visit interaction.



Table 14.2.6.1: Sensitivity Analysis of Primary Endpoints: Absolute Change from Baseline in Lesion Counts and Dichotomized IGA Success at Week 12 (Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Skewness<br>P-Value | Treatment P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count – Absolute Change | | | | |
| from Baseline | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| $LSSD^a$ | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| Non-Inflammatory Lesion Count – Absolute Change<br>from Baseline<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| At Least Two Grade Reduction from Baseline and<br>Achieving Clear or Almost Clear<br>Success<br>Failure | xx.x%<br>xx.x% | xx.x%<br>xx.x% | N/A | $x.xxx^d$ |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (regression model) used to impute missing values.

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset. The average p-value is presented.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Table 14.2.7.1: Sensitivity Tipping-Point Analysis of the Primary Endpoint: Lesion Counts at Week 12 (Intent-to-Treat Population)

| | Lesion Count | Non-Inflammator | y Lesion Count |
|-------------|----------------------|-----------------|----------------------|
| Shift Value | P-Value <sup>a</sup> | Shift Value | P-Value <sup>a</sup> |
| x.xx | X.XXX | X.XX | X.XXX |
| X.XX | X.XXX | X.XX | X.XXX |
| X.XX | x.xxx | X.XX | X.XXX |
| x.xx | X.XXX | X.XX | X.XXX |

<sup>&</sup>lt;sup>a</sup> P-value from an analysis of covariance with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate.

Note: Multiple imputation (MCMC) used to impute missing values, with shift values applied to the imputed lesion count values from E-BPO/E-ATRA 3%/0.1% Cream group. Values have been adjusted for multiple imputation.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

{NOTE TO PROGRAMMER: ADJUST FOOTNOTE "a" TO THE FOLLOWING IF THE NON-PARAMETRIC ANLYSIS WAS CONSIDERED TO BE THE CORRECT ANALYSIS FOR THE PRIMARY EFFICACY ANLYSIS: "P-value from a ranked analysis of covariance with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate."}



Table 14.2.8.1: Secondary Efficacy Analyses
(Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count – Percent Change | (= : :::::) | (= : ::::::) | | |
| from Baseline to Week 12<br>LSMean <sup>a</sup> | VV V | VV V | x.xxx <sup>b</sup> | x.xxx <sup>a</sup> |
| LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | X.XXX | X.XXX<br>X.XXX <sup>c</sup> |
| Loop | ΑΛ.ΑΛ | ΑΛ.ΛΛ | | Λ.ΛΛΛ |
| Non-Inflammatory Lesion Count – Percent Change from Baseline to Week 12 | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| $LSSD^a$ | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| At Least 4-Point Reduction on Item 1 (Pimples) of the PRE-FACE from Baseline to Week 12 Success Failure | xx.x%<br>xx.x% | xx.x%<br>xx.x% | N/A | $x.xxx^d$ |
| At Least 4-Point Reduction on Item 5 (Embarrassment) of the PRE-FACE from Baseline to Week 12 Success Failure | xx.x%<br>xx.x% | xx.x%<br>xx.x% | N/A | $\mathbf{x}.\mathbf{x}\mathbf{x}\mathbf{x}^{\mathrm{d}}$ |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (MCMC) used to impute missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

{NOTE TO PROGRAMMER: ADJUST FOOTNOTE "d" IF FIRTH'S PENALIZED LIKELIHOOD IS NEEDED}

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset. The average p-value is presented.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Table 14.2.8.1: Secondary Efficacy Analyses (Intent-to-Treat Population) 

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count –Absolute Change | | | | |
| from Baseline to Week 8 | | | | |
| LSMeana | XX.X | XX.X | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LSSD <sup>a</sup> | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| Non-Inflammatory Lesion Count -Absolute Change | | | | |
| from Baseline to Week 8 | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | x.xxx <sup>a</sup> |
| LSSD <sup>a</sup> | XX.XX | XX.XX | | x.xxx <sup>c</sup> |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (MCMC) used to impute missing values.

b Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset. The average p-value is presented.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Table 14.2.8.1: Secondary Efficacy Analyses (Intent-to-Treat Population) 

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count – Absolute Change | | | | |
| from Baseline to Week 4 | | | | |
| LSMeana | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| LSSD <sup>a</sup> | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| Non-Inflammatory Lesion Count – Absolute Change from Baseline to Week 4 | | | | |
| | | | b | a |
| LSMean <sup>a</sup> | XX.X | XX.X | X.XXX <sup>b</sup> | X.XXX <sup>a</sup> |
| LSSD <sup>a</sup> | XX.XX | XX.XX | | x.xxx <sup>c</sup> |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (MCMC) used to impute missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Repeat Table 14.2.8.1 for the following table:

Table 14.2.8.2: Secondary Efficacy Analyses (Per-Protocol Population)

Change footnote to "Note: Missing values imputed using last observation carried forward."

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset. The average p-value is presented.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the pimples on your face today <sup>a</sup> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the pimples on your face today <sup>a</sup><br>Week 4 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| n | XX | XX |
| Mean | | |
| | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx.x% | $XX.X^0\!\!/_{\!0}$ |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the pimples on your face today <sup>a</sup> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Week 8 | VV | VV |
| n<br>Mean | XX | XX |
| | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the pimples on your face today <sup>a</sup> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | XX.X% | xx.x% |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1 Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the blackheads on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the blackheads on your face today<br>Week 4 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| | XX | XX |
| n<br>Mean | | |
| SD | XX.X<br>XX.XX | XX.X<br>XX.XX |
| Median | XX.X | XX.XX<br>XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the blackheads on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 8 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the blackheads on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx (xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1 Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the whiteheads on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | , |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = No whiteheads, 10 = Whiteheads as bad as you can imagine



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the whiteheads on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = No whiteheads, 10 = Whiteheads as bad as you can imagine



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the whiteheads on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 8 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = No whiteheads, 10 = Whiteheads as bad as you can imagine



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the whiteheads on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx (xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = No whiteheads, 10 = Whiteheads as bad as you can imagine



Table 14.2.9.1 Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the redness on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the redness on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the redness on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 8 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Rate the redness on your face today | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.9.1 Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how embarrassed you felt because of the acne on your face <sup>a</sup> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not embarrassed at all, 10 = Extremely embarrassed



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how embarrassed you felt because of the acne on your face <sup>a</sup> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not embarrassed at all, 10 = Extremely embarrassed



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how embarrassed you felt because of the acne on your face <sup>a</sup> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 8 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not embarrassed at all, 10 = Extremely embarrassed


Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how embarrassed you felt because of the acne on your face <sup>a</sup> Week 12 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx.x% | xx.x% |
| Failure | xx.x% | xx.x% |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not embarrassed at all, 10 = Extremely embarrassed



Table 14.2.9.1 Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how self-conscious you felt because of the acne on your face. | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx (xx.x%) |
| Failure | xx ( xx.x%) | xx(xx%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not self-conscious at all, 10 = Extremely self-conscious



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how self-conscious you felt because of the acne on your face. | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not self-conscious at all, 10 = Extremely self-conscious



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how self-conscious you felt because of the acne on your face. | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Week 8 | (IV AAA) | (II AAA) |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not self-conscious at all, 10 = Extremely self-conscious



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how self-conscious you felt because of the acne on your face. Week 12 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx (xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not self-conscious at all, 10 = Extremely self-conscious



Table 14.2.9.1 Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how sad you felt because of the acne on your face. | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not sad at all, 10 = Extremely sad



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how sad you felt because of | E-BPO/E-ATRA 3%/0.1% Cream | Vehicle Cream |
|---|---|---|
| the acne on your face. | (N=xxx) | (N=xxx) |
| Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx (xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not sad at all, 10 = Extremely sad



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how sad you felt because of the acne on your face. | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Week 8 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | xx ( xx.x%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not sad at all, 10 = Extremely sad



Table 14.2.9.1: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Intent-to-Treat Population)


| Over the past seven days, rate how sad you felt because of | E-BPO/E-ATRA 3%/0.1% Cream | Vehicle Cream |
|---|---|---|
| the acne on your face. | (N=xxx) | (N=xxx) |
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| At Least 4-Point Reduction from Baseline | | |
| Success | XX (XX.X%) | xx ( xx.x%) |
| Failure | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).

Note: 0 = Not sad at all, 10 = Extremely sad

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.2.9.1 for the following table:

Table 14.2.9.2: Summary of Patient-Reported Evaluation of Facial Acne (PRE-FACE) at Each Evaluation (Per-Protocol Population)

Change footnote to "Last observation carried forward used to impute missing values for only item 1 (pimples) and item 5 (embarrassment).



Table 14.2.10.1: Supportive Efficacy Analyses: PGI-TS, PGI-S, and PGI-C at Week 12 (Intent-to-Treat Population)

| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Treatment<br>P-Value |
|---|---|---|---|
| Patient Global Impression of Treatment Satisfaction (PGI-TS) at Week 12 | | | |
| 0 - I am very satisfied | xx ( xx.x%) | xx ( xx.x%) | $x.xxx^b$ |
| 1 - I am satisfied | xx ( xx.x%) | xx ( xx.x%) | |
| 2 - I am neither satisfied nor dissatisfied | xx ( xx.x%) | xx ( xx.x%) | |
| 3 - I am dissatisfied | xx ( xx.x%) | xx ( xx.x%) | |
| 4 - I am very dissatisfied | xx ( xx.x%) | xx ( xx.x%) | |
| Patient Global Impression of Symptom Severity (PGI-S) at Week 12 | | | |
| 0 - None: no pimples, clear skin | xx ( xx.x%) | xx ( xx.x%) | $x.xxx^b$ |
| 1 - Mild: very few pimples, almost clear skin | xx ( xx.x%) | xx ( xx.x%) | |
| 2 - Moderate: some pimples | xx ( xx.x%) | xx ( xx.x%) | |
| 3 - Severe: many pimples, almost no clear skin | xx ( xx.x%) | xx ( xx.x%) | |
| 4 - Very severe: Large amount of pimples, no clear skin | xx ( xx.x%) | xx ( xx.x%) | |
| At Least "Minimally Improved" in PGI-C from Baseline to Week 12 | | | |
| Success | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> | X.XXX <sup>a</sup> |
| Failure | xx.x% | XX.X% | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

{NOTE TO PROGRAMMER: ADJUST FOOTNOTE "d" IF FIRTH'S PENALIZED LIKELIHOOD IS NEEDED}

P-value from a logistic regression with factors of treatment group and analysis center.
 P-value from a cumulative logistic regression with factors of treatment group and analysis center.



Table 14.2.11.1: Supportive Efficacy Analyses: Lesion Count and IGA (Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| At Least Two Grade Reduction from Baseline and | | | | |
| Achieving Clear or Almost Clear at Week 8 | | | | |
| Success | xx.x% | xx.x% | N/A | $x.xxx^d$ |
| Failure | XX.X% | xx.x% | | |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (MCMC) used to impute missing values.

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Table 14.2.11.1: Supportive Efficacy Analyses: Lesion Count and IGA (Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| At Least Two Grade Reduction from Baseline and | | | | |
| Achieving Clear or Almost Clear at Week 4 | | | | |
| Success | xx.x% | xx.x% | N/A | $x.xxx^d$ |
| Failure | XX.X% | xx.x% | | |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (MCMC) used to impute missing values.

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Table 14.2.11.1: Supportive Efficacy Analyses: Lesion Count and IGA (Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| Inflammatory Lesion Count -Absolute Change | - · | | _ | |
| from Baseline to Week 2 | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| $\mathrm{LSSD^a}$ | XX.XX | xx.xx | | x.xxx <sup>c</sup> |
| Non-Inflammatory Lesion Count –Absolute Change<br>from Baseline to Week 2<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| At Least Two Grade Reduction from Baseline and<br>Achieving Clear or Almost Clear at Week 2<br>Success<br>Failure | xx.x%<br>xx.x% | xx.x%<br>xx.x% | N/A | x.xxx <sup>d</sup> |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

Note: Multiple imputation (MCMC) used to impute missing values.

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> P-value from a logistic regression with factors of treatment group and analysis center.



Table 14.2.12.1: Supportive Efficacy Analyses: PRE-FACE ASD Scores (Intent-to-Treat Population)


| E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|
| · | · | | |
| | | , | |
| XX.X | XX.X | X.XXX <sup>b</sup> | X.XXX <sup>a</sup> |
| XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| XX.X | XX.X | $x.xxx^b$ | x.xxx <sup>a</sup> |
| XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| XX.X | XX.X | $x.xxx^b$ | x.xxx <sup>a</sup> |
| XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| | 3%/0.1% Cream (N=xxx) xx.x xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx | 3%/0.1% Cream (N=xxx) Vehicle Cream (N=xxx) xx.x xx.x xx.xx xx.xx xx.xx xx.xx | 3%/0.1% Cream Vehicle Cream Skewness P-Value xx.x xx.x xx.x xx.xx xx.xx xx.xx |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

b Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> Multiple imputation used to impute missing values for only item 1 (pimples).



Table 14.2.12.1: Supportive Efficacy Analyses: PRE-FACE ASD Scores (Intent-to-Treat Population)


| (N=xxx) | P-Value | Treatment<br>P-Value |
|---|---|---|
| | , | |
| XX.X | X.XXX <sup>b</sup> | X.XXX <sup>a</sup> |
| XX.XX | | x.xxx <sup>c</sup> |
| XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| XX.XX | | x.xxx <sup>c</sup> |
| XX.X | $x.xxx^b$ | x.xxx <sup>a</sup> |
| XX.XX | | x.xxx <sup>c</sup> |
| XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| XX.XX | | x.xxx <sup>c</sup> |
| | XX.XX XX.XX XX.XX XX.XX | XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

b Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> Multiple imputation used to impute missing values for only item 1 (pimples).



Table 14.2.12.1: Supportive Efficacy Analyses: PRE-FACE ASD Scores (Intent-to-Treat Population)


| E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|
| (= : :::::) | | | |
| XX.X | XX.X | $x.xxx^b$ | $\mathbf{X}.\mathbf{X}\mathbf{X}\mathbf{X}^{\mathbf{a}}$ |
| XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| xx.x | xx.x | x.xxx <sup>b</sup> | X.XXX <sup>a</sup> |
| XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| | 3%/0.1% Cream (N=xxx) xx.x xx.xx xx.x xx.xx xx.xx xx.xx | 3%/0.1% Cream (N=xxx) Vehicle Cream (N=xxx) xx.x xx.x xx.xx xx.xx xx.xx xx.xx | 3%/0.1% Cream Vehicle Cream Skewness P-Value xx.x xx.x xx.x xx.xx xx.xx xx.xx |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

b Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> Multiple imputation used to impute missing values for only item 1 (pimples).



Table 14.2.13.1: Supportive Efficacy Analyses: PRE-FACE AID Scores (Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment P-Value |
|---|---|---|---|---|
| PRE-FACE Item 5 (Embarrassed) –Absolute Change | | | | |
| from Baseline to Week 8 <sup>d</sup> | | | | |
| LSMeana | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| $\mathrm{LSSD}^{\mathrm{a}}$ | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| PRE-FACE Item 6 (Self-Conscious) –Absolute<br>Change from Baseline to Week 8<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| PRE-FACE Item 7 (Sad) –Absolute Change<br>from Baseline to Week 8<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

b Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

<sup>&</sup>lt;sup>d</sup> Multiple imputation used to impute missing values for only item 5 (embarrassed).



Table 14.2.13.1: Supportive Efficacy Analyses: PRE-FACE AID Scores (Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| PRE-FACE Item 5 (Embarrassed) –Absolute Change | | | | |
| from Baseline to Week 4 <sup>d</sup> | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| $LSSD^a$ | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| PRE-FACE Item 6 (Self-Conscious) –Absolute<br>Change from Baseline to Week 4<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| PRE-FACE Item 7 (Sad) –Absolute Change<br>from Baseline to Week 4<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

<sup>&</sup>lt;sup>b</sup> Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

d Multiple imputation used to impute missing values for only item 5 (embarrassed).



Table 14.2.13.1: Supportive Efficacy Analyses: PRE-FACE AID Scores (Intent-to-Treat Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | Skewness<br>P-Value | Treatment<br>P-Value |
|---|---|---|---|---|
| PRE-FACE Item 5 (Embarrassed) – Absolute Change | | | | |
| from Baseline to Week 2 <sup>d</sup> | | | | |
| LSMean <sup>a</sup> | XX.X | XX.X | $x.xxx^b$ | X.XXX <sup>a</sup> |
| $LSSD^a$ | XX.XX | XX.XX | | x.xxx <sup>c</sup> |
| PRE-FACE Item 6 (Self-Conscious) –Absolute<br>Change<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | x.xxx <sup>b</sup> | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |
| PRE-FACE Item 7 (Sad) –Absolute Change<br>from Baseline to Week 2<br>LSMean <sup>a</sup><br>LSSD <sup>a</sup> | XX.X<br>XX.XX | XX.X<br>XX.XX | $x.xxx^b$ | X.XXX <sup>a</sup><br>X.XXX <sup>c</sup> |

<sup>&</sup>lt;sup>a</sup> Least squares means, standard deviations and treatment p-value from an analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.

b Skewness test, based on methods presented by J.H. Zar (1984), assessed for each imputed dataset.

<sup>&</sup>lt;sup>c</sup> P-value from a ranked analysis of covariance with factors of treatment and analysis center and the respective Baseline lesion count as a covariate.

d Multiple imputation used to impute missing values for only item 5 (embarrassed).



Table 14.2.14.1: Summary of Patient Global Impression of Change (PGI-C) at Each Evaluation (Intent-to-Treat Population)


| Since the start of the study, how have your acne symptoms changed? Week 2 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| n | XX | XX |
| 0 - Very much improved | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Much improved | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Minimally improved | xx ( xx.x%) | xx ( xx.x%) |
| 3 - No Change | xx (xx.x%) | xx ( xx.x%) |
| 4 - Minimally worse | xx ( xx.x%) | xx ( xx.x%) |
| 5 - Much worse | xx ( xx.x%) | xx ( xx.x%) |
| 6 - Very much worse | xx ( xx.x%) | xx ( xx.x%) |
| At least minimally improved | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0 - Very much improved | xx ( xx.x%) | xx (xx.x%) |
| 1 - Much improved | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Minimally improved | xx ( xx.x%) | xx (xx.x%) |
| 3 - No Change | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Minimally worse | xx ( xx.x%) | xx ( xx.x%) |
| 5 - Much worse | xx ( xx.x%) | xx ( xx.x%) |
| 6 - Very much worse | xx ( xx.x%) | xx ( xx.x%) |
| At least minimally improved | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing values. At least minimally improved defined as "very much improved", "much improved", or "minimally improved".



Table 14.2.14.1: Summary of Patient Global Impression of Change (PGI-C) at Each Evaluation (Intent-to-Treat Population)


| Since the start of the study, how have your acne symptoms changed? Week 8 | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| | VV | VV |
| n<br>0 - Very much improved | XX | XX |
| | xx ( xx.x%) | XX ( XX.X%) |
| 1 - Much improved | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Minimally improved | xx ( xx.x%) | xx ( xx.x%) |
| 3 - No Change | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Minimally worse | xx ( xx.x%) | xx ( xx.x%) |
| 5 - Much worse | xx ( xx.x%) | XX (XX.X%) |
| 6 - Very much worse | xx ( xx.x%) | xx ( xx.x%) |
| At least minimally improved | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - Very much improved | xx (xx.x%) | xx ( xx.x%) |
| 1 - Much improved | xx (xx.x%) | xx ( xx.x%) |
| 2 - Minimally improved | xx (xx.x%) | xx ( xx.x%) |
| 3 - No Change | $xx(x^{0})$ | xx ( xx.x%) |
| 4 - Minimally worse | xx ( xx.x%) | xx ( xx.x%) |
| 5 - Much worse | xx ( xx.x%) | xx ( xx.x%) |
| 6 - Very much worse | xx ( xx.x%) | xx ( xx.x%) |
| At least minimally improved | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing values. At least minimally improved defined as "very much improved", "much improved", or "minimally improved".



Table 14.2.15.1: Summary of Patient Global Impression of Symptom Severity (PGI-S) at Each Evaluation (Intent-to-Treat Population)


| Right now, my acne symptoms are: Baseline | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| n | XX | XX |
| 0 - None: no pimples, clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild: very few pimples, almost clear skin | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate: some pimples | xx ( xx.x%) | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}\mathbf{x}\mathbf{x})$ |
| 3 – Severe: many pimples, almost no clear skin | XX (XX.X/0)<br>XX (XX.X%) | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}\mathbf{x}\mathbf{x})$ |
| 4 – Very severe: Large amount of pimples, no clear skin | $\mathbf{x}\mathbf{x} \ (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}\mathbf{x}\mathbf{x}')$ |
| 4 - Very severe. Large amount of pumples, no clear skin | AA ( AA.A/0) | AA ( AA.A/0) |
| Week 2 | | |
| n | XX | XX |
| 0 - None: no pimples, clear skin | $XX (XX.X^{0})$ | xx (xx.x%) |
| 1 – Mild: very few pimples, almost clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate: some pimples | xx ( xx.x%) | xx (xx.x%) |
| 3 – Severe: many pimples, almost no clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Very severe: Large amount of pimples, no clear skin | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0 - None: no pimples, clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild: very few pimples, almost clear skin | XX (XX.X/0)<br>XX (XX.X%) | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}\mathbf{x}\mathbf{x})$ |
| 2 – Moderate: some pimples | XX (XX.X/0)<br>XX (XX.X%) | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}^{\prime\prime})$ |
| 3 – Severe: many pimples, almost no clear skin | | xx ( xx.x%) |
| 4 – Very severe: Large amount of pimples, no clear skin | | |
| 4 – very severe: Large amount of pimples, no clear skin | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.15.1: Summary of Patient Global Impression of Symptom Severity (PGI-S) at Each Evaluation (Intent-to-Treat Population)


| Right now, my acne symptoms are: | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 8 | | |
| n | XX | XX |
| 0 - None: no pimples, clear skin | XX (XX.X%) | XX (XX.X%) |
| 1 – Mild: very few pimples, almost clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate: some pimples | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe: many pimples, almost no clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Very severe: Large amount of pimples, no clear skin | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None: no pimples, clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild: very few pimples, almost clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate: some pimples | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe: many pimples, almost no clear skin | xx ( xx.x%) | xx ( xx.x%) |
| 4 – Very severe: Large amount of pimples, no clear skin | xx ( xx.x%) | xx ( xx.x%) |



Table 14.2.16.1: Summary of Patient Global Impression of Treatments Satisfaction (PGI-TS) at Each Evaluation (Intent-to-Treat Population)


| Right now, how satisfied are you with your acne treatment: | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 2 | | |
| n | XX | XX |
| 0 – I am very satisfied | xx ( xx.x%) | xx (xx.x%) |
| 1 – I am satisfied | xx (xx.x%) | xx (xx.x%) |
| 2 – I am neither satisfied not dissatisfied | xx (xx.x%) | xx (xx.x%) |
| 3 – I am dissatisfied | xx (xx.x%) | xx ( xx.x%) |
| 4 – I am very dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0 – I am very satisfied | xx ( xx.x%) | xx ( xx.x%) |
| 1 – I am satisfied | xx ( xx.x%) | xx (xx.x%) |
| 2 – I am neither satisfied not dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| 3 – I am dissatisfied | xx (xx.x%) | xx (xx.x%) |
| 4 – I am very dissatisfied | XX (XX.X%) | xx ( xx.x%) |



Table 14.2.16.1: Summary of Patient Global Impression of Treatments Satisfaction (PGI-TS) at Each Evaluation (Intent-to-Treat Population)


| Right now, how satisfied are you with your acne treatment: | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Week 8 | | |
| n | XX | XX |
| 0 – I am very satisfied | xx ( xx.x%) | xx ( xx.x%) |
| 1 – I am satisfied | xx ( xx.x%) | xx ( xx.x%) |
| 2 – I am neither satisfied not dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| 3 – I am dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| 4 – I am very dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 – I am very satisfied | xx ( xx.x%) | xx ( xx.x%) |
| 1 – I am satisfied | xx ( xx.x%) | xx ( xx.x%) |
| 2 – I am neither satisfied not dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| 3 – I am dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| 4 – I am very dissatisfied | xx ( xx.x%) | xx ( xx.x%) |
| | • | |



Table 14.2.17.1: Summary of Acne-QoL Questionnaire Responses at Baseline and Week 12 (Intent-to-Treat Population)


| Self-Perception Domain | E-BPO/E-ATRA 3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | xx.xx |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Self-Perception domain calculated from the questions 1, 2, 3, 6, and 10.

Role-Emotional domain calculated from questions 4, 5, 7, 8, and 9.

Role-Social domain calculated from questions 11, 12, 13, and 14.

Acne Symptoms domain calculated from questions 15, 16, 17, 18, and 19.



Table 14.2.17.1: Summary of Acne-QoL Questionnaire Responses at Baseline and Week 12 (Intent-to-Treat Population)


| Role-Emotional Domain | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Self-Perception domain calculated from the questions 1, 2, 3, 6, and 10.

Role-Emotional domain calculated from questions 4, 5, 7, 8, and 9.

Role-Social domain calculated from questions 11, 12, 13, and 14.

 $Acne \ Symptoms \ domain \ calculated \ from \ questions \ 15, \ 16, \ 17, \ 18, \ and \ 19.$ 



Table 14.2.17.1: Summary of Acne-QoL Questionnaire Responses at Baseline and Week 12 (Intent-to-Treat Population)


| Role-Social Domain | E-BPO/E-ATRA 3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Self-Perception domain calculated from the questions 1, 2, 3, 6, and 10.

Role-Emotional domain calculated from questions 4, 5, 7, 8, and 9.

Role-Social domain calculated from questions 11, 12, 13, and 14.

Acne Symptoms domain calculated from questions 15, 16, 17, 18, and 19.



Table 14.2.17.1: Summary of Acne-QoL Questionnaire Responses at Baseline and Week 12 (Intent-to-Treat Population)


| Acne Symptoms Domain | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Absolute Change from Baseline | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |

Self-Perception domain calculated from the questions 1, 2, 3, 6, and 10.

Role-Emotional domain calculated from questions 4, 5, 7, 8, and 9.

Role-Social domain calculated from questions 11, 12, 13, and 14.

Acne Symptoms domain calculated from questions 15, 16, 17, 18, and 19.



Table 14.3.0.1: Summary of Extent of Exposure (Safety Population)

| | E-BPO/E-ATRA 3%/0.1% Cream | Vehicle Cream |
|---|---|---|
| | (N=xxx) | (N=xxx) |
| Fotal Number of Days of Exposure | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Fotal Number of Applications | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Fotal Number of Missed Applications | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Compliant <sup>a</sup> | | |
| n | XX | XX |
| Yes | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> A subject was considered compliant with the dosing regimen if the subject applied 80-120% of the expected number of applications and did not miss more than 5 consecutive applications while enrolled in the study.



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Erythema | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|--------------|------------------------------------|--------------------------|
| Baseline | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | XX ( XX.X%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Erythema | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|--------------|------------------------------------|-----------------------|
| Week 8 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx(xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx(xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx(xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Scaling | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|--------------|------------------------------------|--------------------------|
| Baseline | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx (xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Scaling | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|--------------|------------------------------------|-----------------------|
| Week 8 | | |
| n | XX | XX |
| 0 - None | XX ( XX.X%) | xx (xx.x%) |
| 1 - Mild | xx(xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx(xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx(xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx(xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Pigmentation | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|--------------|------------------------------------|--------------------------|
| Baseline | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Pigmentation | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|--------------|------------------------------------|--------------------------|
| Week 8 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx (xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx(xx.x%) | xx ( xx.x%) |
| 2 – Moderate | $xx(xx.x^{0})$ | xx ( xx.x%) |
| 3 – Severe | $xx(xx.x^{0})$ | xx ( xx.x%) |


Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Dryness | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| 0-None | xx (xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| 0-None | xx (xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0-None | xx (xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx (xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Dryness | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|--------------|------------------------------------|--------------------------|
| Week 8 | | |
| n | XX | XX |
| 0 - None | xx (xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx (xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None | xx (xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx(xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Itching | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|--------------|------------------------------------|--------------------------|
| Baseline | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx (xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Itching | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|--------------|------------------------------------|-----------------------|
| Week 8 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 - Mild | xx (xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx(xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Burning | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|--------------|------------------------------------|--------------------------|
| Baseline | | |
| n | XX | XX |
| 0-None | xx (xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| 0-None | xx (xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Burning | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|--------------|------------------------------------|-----------------------|
| Week 8 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx(xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx(xx.x%) | xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Stinging | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 2 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0-None | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Mild | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild<br>2 – Moderate | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |



Table 14.3.1.1: Summary of Cutaneous Signs and Local Tolerability at Each Evaluation (Safety Population)


| Stinging | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|--------------|------------------------------------|-----------------------|
| Week 8 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx(xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx(xx.x%) | xx ( xx.x%) |



Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| Subjects Reporting Any Treatment-Emergent Adverse Event Number of Treatment-Emergent Adverse Events | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx)<br>xx (xx.x%)<br>xx | Vehicle Cream (N=xxx) xx (xx.x%) xx |
|---|---|---|
| Subjects Reporting Any Serious Treatment-Emergent Adverse Event<br>Number of Serious Treatment-Emergent Adverse Events | xx ( xx.x%)<br>xx | xx ( xx.x%)<br>xx |
| Subjects Reporting Treatment-Emergent Adverse Event with Outcome of Fatal Number of Treatment-Emergent Adverse Events with Outcome of Fatal | xx ( xx.x%)<br>xx | xx ( xx.x%)<br>xx |
| Subjects Who Discontinued Study Drug Due to a Treatment-Emergent Adverse Event<br>Number of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug | xx ( xx.x%)<br>xx | xx ( xx.x%)<br>xx |
| Subjects Who Discontinued from the Study Due to a Treatment-Emergent Adverse Event Number of Treatment-Emergent Adverse Events Leading to Discontinuation of Study | xx (xx.x%)<br>xx | xx (xx.x%)<br>xx |

Note: Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)


| | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| By Maximum Severity | | |
| Severe | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) |
| By Strongest Relationship to Study Drug | | |
| Related | XX (XX.X%) | xx ( xx.x%) |
| Not Related | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity within Relationship to Study Drug | | |
| Related | | |
| Severe | XX (XX.X%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) |
| Not Related | , , | , , |
| Severe | XX (XX.X%) | xx ( xx.x%) |
| Moderate | xx ( xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.2.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) | P-Value <sup>b</sup> |
|---|---|---|---|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx ( xx.x%) | xx ( xx.x%) | X.XXX |
| | xx ( xx.x%) | xx ( xx.x%) | X.XXX |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application.

b P-value for the difference between treatment groups from a Fisher's Exact test. The specific system organ classes and preferred terms analyzed will be those that are reported by at least one percent of the patients in any treatment group.



Table 14.3.1.2.3: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | <u>Severity</u> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxx | Severe | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) |
| | Mild | xx ( xx.x%) | xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Severe | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) |
| | Mild | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported reported severity.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application.



Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Relationship to Study Drug (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | <u>Relationship</u> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxx | Related | xx ( xx.x%) | xx ( xx.x%) |
| | Not Related | xx ( xx.x%) | xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxx | Related | xx ( xx.x%) | xx ( xx.x%) |
| | Not Related | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| Subjects Reporting Any Serious Treatment-Emergent Adverse Event Number of Serious Treatment-Emergent Adverse Events | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) xx (xx.x%) xx | Vehicle Cream (N=xxx) xx (xx.x%) xx |
|---|---|---|
| Subjects Reporting Serious Treatment-Emergent Adverse Event with Outcome of Fatal Number of Serious Treatment-Emergent Adverse Events with Outcome of Fatal | xx ( xx.x%)<br>xx | xx (xx.x%) |
| Subjects Who Discontinued Study Drug Due to a Serious Treatment-Emergent Adverse Event Number of Serious Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug | xx ( xx.x%)<br>xx | xx (xx.x%)<br>xx |
| Subjects Who Discontinued from the Study Due to a Serious Treatment-Emergent Adverse Event Number of Serious Treatment-Emergent Adverse Events Leading to Discontinuation of Study | xx (xx.x%)<br>xx | xx (xx.x%)<br>xx |

Note: Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| By Maximum Severity | | |
| Severe | XX (XX.X%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) |
| By Strongest Relationship to Study Drug | | |
| Related | xx (xx.x%) | xx ( xx.x%) |
| Not Related | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity within Relationship to Study Drug | | |
| Related | | |
| Severe | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) |
| Mild | xx (xx.x%) | xx ( xx.x%) |
| Not Related | | ` ' |
| Severe | xx (xx.x%) | xx ( xx.x%) |
| Moderate | xx (xx.x%) | xx ( xx.x%) |
| Mild | xx ( xx.x%) | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.3.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)


| System Organ Class <sup>a</sup> Preferred Term | E-BPO/E-ATRA<br>3%/0.1% Cream<br>(N=xxx) | Vehicle Cream (N=xxx) | P-Value <sup>b</sup> |
|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xx ( xx.x%) | xx ( xx.x%) | x.xxx |
| | xx ( xx.x%) | xx ( xx.x%) | x.xxx |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: MedDRA Version 21.0

Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application.

b P-value for the difference between treatment groups from a Fisher's Exact test. The specific system organ classes and preferred terms analyzed will be those that are reported by at least one percent of the patients in any treatment group.



Table 14.3.1.3.3: Summary of Serious Treatment-Emergent Adverse Events by Severity (Safety Population)


| System Organ Class <sup>a</sup> <u>Preferred Term</u> | Severity _ | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxx | Severe | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) |
| | Mild | xx ( xx.x%) | xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxxx | Severe | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) |
| | Mild | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application.



Table 14.3.1.3.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship to Study Drug (Safety Population)

| System Organ Class <sup>a</sup> Preferred Term | <u>Relationship</u> | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|---|
| xxxxxxxxxxxxxxxxxxxxxx | Related | xx ( xx.x%) | xx ( xx.x%) |
| | Not Related | xx ( xx.x%) | xx ( xx.x%) |
| xxxxxxxxxxxxxxxxxxxxxxx | Related | xx ( xx.x%) | xx ( xx.x%) |
| | Not Related | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: MedDRA Version 21.0.

Treatment-emergent adverse events are those events that were not indicated as occurring prior to first application. Related defined as "Definitely", "Probably", or "Possible". Not Related defined as "Unlikely" or "Not related".



Table 14.3.1.4: Summary of Vital Signs (Safety Population)


| Temperature (°C) | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.3.1.4: Summary of Vital Signs (Safety Population)


| Respiratory Rate (breaths/min) | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | (IV ANA) | (IV AAA) |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.3.1.4: Summary of Vital Signs (Safety Population) 

| Systolic Blood Pressure (mmHg) | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.3.1.4: Summary of Vital Signs (Safety Population)


| Diastolic Blood Pressure (mmHg) | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.3.1.4: Summary of Vital Signs (Safety Population)


| Heart Rate (beats/min) | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Week 12 | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx |



Table 14.3.1.4.2: Shift Table of Vital Signs (Safety Population)

| | E-BPC | D/E-ATRA 3%/0.1%<br>(N=xxx) | 6 Cream | | Vehicle Cream<br>(N=xxx) | |
|---|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | | Week 12 | | | Week 12 | |
| Baseline | <90 mmHg | 90-140 mmHg | >140 mmHg | <90 mmHg | 90-140 mmHg | >140 mmHg |
| <90 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90-140 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >140 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Diastolic Blood Pressure (mmHg) | | Week 12 | | | Week 12 | |
| <u>Baseline</u> | <90 mmHg | 90-100 mmHg | >100 mmHg | <90 mmHg | 90-100 mmHg | >100 mmHg |
| <90 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 90-100 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >100 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Heart Rate (beats/min) | | Week 12 | | | Week 12 | |
| Baseline | <60 bpm | 60-100 bpm | >100 bpm | <60 bpm | 60-100 bpm | >100 bpm |
| <60 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 60-100 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >100 mmHg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.5: Summary of Abnormal Physical Examination Findings by Visit (Safety Population)

| | E-BPO 3% Cream | Vehicle Cream |
|---|---|---|
| | $\underline{\hspace{1cm}(N=xxx)}$ | (N=xxx) |
| Heart<br>Baseline | | |
| n | XX | XX |
| Abnormal | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| Abnormal | xx ( xx.x%) | xx ( xx.x%) |
| Lung<br>Baseline | | |
| n | XX | XX |
| Abnormal | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| Abnormal | xx ( xx.x%) | xx ( xx.x%) |
| <b>Abdomen</b><br>Baseline | | |
| n | XX | XX |
| Abnormal | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | |
| n | XX | XX |
| Abnormal | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.6: Summary of Patient Global Impression of Treatment Side-Effects (PGI-SE) at Each Evaluation (Safety Population)


| Right now, how bothered are you by the side effects of your acne treatment: | E-BPO/E-ATRA 3%/0.1% Cream (N=xxx) | Vehicle Cream (N=xxx) |
|---|---|---|
| Week 2 | | |
| n | XX | XX |
| 0 - I am not bothered | xx ( xx.x%) | xx ( xx.x%) |
| 1 - I am somewhat bothered | xx ( xx.x%) | xx ( xx.x%) |
| 2 - I am moderately bothered | xx ( xx.x%) | xx ( xx.x%) |
| 3 - I am very bothered | xx ( xx.x%) | xx ( xx.x%) |
| 4 - I am extremely bothered | xx ( xx.x%) | xx ( xx.x%) |
| Week 4 | | |
| n | XX | XX |
| 0 - I am not bothered | xx ( xx.x%) | xx ( xx.x%) |
| 1 - I am somewhat bothered | xx ( xx.x%) | xx ( xx.x%) |
| 2 - I am moderately bothered | xx ( xx.x%) | xx ( xx.x%) |
| 3 - I am very bothered | xx ( xx.x%) | xx ( xx.x%) |
| 4 - I am extremely bothered | xx ( xx.x%) | xx ( xx.x%) |
| Week 8 | | |
| n | XX | XX |
| 0 - I am not bothered | xx ( xx.x%) | xx ( xx.x%) |
| 1 - I am somewhat bothered | xx ( xx.x%) | xx ( xx.x%) |
| 2 - I am moderately bothered | xx ( xx.x%) | xx ( xx.x%) |
| 3 - I am very bothered | xx ( xx.x%) | xx ( xx.x%) |
| 4 - I am extremely bothered | xx ( xx.x%) | xx ( xx.x%) |



Table 14.3.1.6: Summary of Patient Global Impression of Treatment Side-Effects (PGI-SE) at Each Evaluation (Safety Population)


| Right now, how bothered are you by the side effects of your acne treatment: | E-BPO/E-ATRA 3%/0.1% Cream<br>(N=xxx) | Vehicle Cream<br>(N=xxx) |
|---|---|---|
| Week 12 | | |
| n | XX | XX |
| 0 - I am not bothered | xx (xx.x%) | xx (xx.x%) |
| 1 - I am somewhat bothered | xx ( xx.x%) | xx ( xx.x%) |
| 2 - I am moderately bothered | xx ( xx.x%) | xx (xx.x%) |
| 3 - I am very bothered | xx ( xx.x%) | xx ( xx.x%) |
| 4 - I am extremely bothered | xx (xx.x%) | xx (xx.x%) |



### 13. INDEX OF PLANNED FIGURES

| Figure 14.2.7.2: Sensiti | vity Tipping-Poin | t Analysis of the | Primary Endpoint | : Treatment Success |
|---|---|---|---|---|
| | in IGA at Week | 12 (Intent-to-T | reat Population) | 173 |



Figure 14.2.7.2: Sensitivity Tipping-Point Analysis of the Primary Endpoint: Treatment Success in IGA at Week 12 (Intent-to-Treat Population)



Note: The horizontal and vertical axes indicate the number of successes that can potentially be observed among nonrespondents in the each treatment group. Each plotted point indicates the number of imputed successes in each treatment group that would alter the study's conclusion with the staircase region indicating the tipping points of the study.

The red lines represent average number of imputed successes from the primary analysis using multiple imputation (MCMC) to impute missing values.



### 14. INDEX OF PLANNED LISTINGS

| Listing 16.1.7: Randomization Scheme | 176 |
|---|---|
| Listing 16.2.1.1: End of Study Information | 177 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria | 178 |
| Listing 16.2.2.2: Screen Failure | 179 |
| Listing 16.2.2.3: Protocol Deviations | 180 |
| Listing 16.2.3: Analysis Populations | 181 |
| Listing 16.2.4.1: Subject Demographic Information | 182 |
| Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Cl<br>and Preferred Terms | |
| Listing 16.2.4.2.2: Medical/Surgical History | 184 |
| Listing 16.2.4.3.1: Unique Medication Names Coded to WHO Drug Global Dictionary AT Level 2 Terms and Preferred Names | |
| Listing 16.2.4.3.2: Prior and Concomitant Medications | 186 |
| Listing 16.2.4.4.1: Unique Procedure/Therapy Names Coded to MedDRA System Organ C and Preferred Terms | |
| Listing 16.2.4.4.2: Prior and Concomitant Procedures/Therapies | 188 |
| Listing 16.2.5.1: Study Visit Compliance | 189 |
| Listing 16.2.5.2: Subject Dosing Compliance | 190 |
| Listing 16.2.5.3: Subject Dosing Deviations | 191 |
| Listing 16.2.5.4: Study Medication Accountability Log | 192 |
| Listing 16.2.5.5: Photography | 193 |
| Listing 16.2.6.1: Investigator Global Assessment | 194 |
| Listing 16.2.6.2: Lesion Counts | 195 |
| Listing 16.2.6.3.1: Acne-QoL Descriptions | 196 |
| Listing 16.2.6.3.2: Acne-QoL | 198 |
| Listing 16.2.6.3.3: Acne-QoL Domain Scores | 199 |
| Listing 16.2.6.4: PRO - Patient Reported Evaluation of Facial Acne (PRE-FACE) | 200 |
| Listing 16.2.6.5: PRO - Patient Reported Impression of Symptom Severity (PGI-S) | 201 |
| Listing 16.2.6.6: PRO – Patient Global Impression of Change (PGI-C), Patient Global Impression of Treatment Satisfaction (PGI-TS), Patient Global Impression of Treatment Side-Effects (PGI-SE) | 202 |

TOOL.AN.10-01.01 Statistical Analysis Plan



| Listing 16.2.7.1: Cutaneous Signs and Local Tolerability | 203 |
|---|---|
| Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms | 204 |
| Listing 16.2.7.2.2: Pre-Treatment Adverse Events | 205 |
| Listing 16.2.7.2.3: Treatment-Emergent Adverse Events | 206 |
| Listing 16.2.7.2.4: Serious Adverse Events | 207 |
| Listing 16.2.7.2.5: Subjects Who Prematurely Discontinued Study and/or Discontinued Study Drug Due to Adverse Events | • |
| Listing 16.2.8.1: Urine Pregnancy Tests | 209 |
| Listing 16.2.8.2: Physical Examination | 210 |
| Listing 16.2.8.3: Vital Signs | 211 |



## Listing 16.1.7: Randomization Scheme (Page xx of yy)

| Subject | Age/Sex | Eval | Randomization Date | Kit Number | Assigned Arm |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | xxxx | xxxxx xx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | XXXX | xxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | XXXX | xxxxx xx xxxxx |
| XXXXXX | xxxx | xxxxxxxx | xxxxxxxxxxxx | XXXX | xxxxx xx xxxxx |
| XXXXXX | xxxx | xxxxxxxx | xxxxxxxxxxxx | XXXX | xxxxx xx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxx | XXXX | xxxxxxx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxxx | xxxx | xxxxx xx xxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxxxxxxxx | XXXX | xxxxxxx xxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.



## Listing 16.2.1.1: End of Study Information Treatment Arm (Page xx of yy)

Date of Study Continue to the Completion/ Did Subject Date of First Date of Last Discontinuation Complete the Long Term Primary Reason Subject Age/Sex Eval Application Application (Day) 1 the Study for Study Discontinuation Safety Study XXXXXX XXXX XXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXXXXXX XXX X XXX XXXXXXX XXXX XXXXXXX XXXXXX XXXX XXXXXXXX XXXXXXXX xxxxxxxxxx XXXXXXXXXXXX xxxxxxx xxxxx XX X XXX XXXXXXX XXXX XXX XXXXXXX XXXXXX XXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXXXXXXX XX XXXX XX XXXXXXXXX XXX XXXXXXX XXXXX XXXXX XXXXX XXX

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

#### Listing sorted by Subject.

If Primary Reason for Study Discontinuation is Lost to Follow-Up, Protocol Violation, Withdrawal by Subject, or Other, the reason specification will be included following a colon (for example, WITHDRAWAL BY SUBJECT: xxxxx)

If subject will not continue to the LTS, the reason specification will be included in the final column following a colon.

<sup>1</sup> Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



# Listing 16.2.2.1: Inclusion/Exclusion Criteria Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Criterion Failed | Description |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | xxxxxx | xxxxx xxx xx xxxxxxx xxxx xxxx xxxxxxxx |
| xxxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ******* **** *********** |
| xxxxx | xxxx | xxxxxxxx | xxxxx | ***** *** ** ******* **** *********** |
| | | | xxxxx | ***** *** ** ******* **** *********** |
| | | | xxxxx | xxxxx xxx xx xxxxxxx xxxx xxxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Criterion Failed.



## Listing 16.2.2.2: Screen Failure (Page xx of yy)

| Subject | Age/Sex | Eval | Date of<br>Screen Failure | Reason for Screen Failure |
|---|---|---|---|---|
| xxx | xxxx | xxxxxxxx | xxxxxxxxx | ***** *** ** ******* *** ************* |
| xx | xxxx | xxxxxxxx | xxxxxxxxx | ***** *** ** ******* **** ************* |
| X | xxxx | xxxxxxxx | xxxxxxxxx | ***** *** ** ******* *** ************** |
| | | | xxxxxxxxx | ***** *** ** ******* *** ************** |
| | | | xxxxxxxxx | ***** *** ** ******* *** ************ **** |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.



# Listing 16.2.2.3: Protocol Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Deviation | Date (Day <sup>1</sup> ) |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx | ****** * ******* *** ** ****** *** *** *** *** *** | xxxxxxxxxxxx |
| | | | xxxxxx xxx xx xxxxxx xxxxxx xxx xxx xx | xxxxxxxxxxxx |
| | | | xxxxxx x xxxxxxxx | |
| xxxxxx | XXXX | xxxxxxxx | XXXXXX XXX XX XXXXXX XXXXXX XXX XXX XX | xxxxxxxxxxxx |
| xxxxx | xxxx | xxxxxxxx | xxxxxx xxx xx xxxxxx xxxxxx xxx xxx xx | xxxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Date.

<sup>1</sup> Day is calculated as date - Baseline date for dates prior to Baseline visit. Otherwise, day is calculated as date - Baseline date + 1 for dates on or after Baseline visit.


# Listing 16.2.3: Analysis Populations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Population | Included Reason(s) Excluded | Exception(s) |
|---|---|---|---|---|
| xxxxx | xxxx | Intent-to-Treat<br>Safety<br>Per-Protocol | xxx<br>xx xxxxxxxxx xxxxxxx xxxxxxxx<br>xx xxxxxx | |
| xxxxxx | xxxx | Intent-to-Treat<br>Safety<br>Per-Protocol | xxx<br>xxx<br>xxx | ******* |
| xxxxx | xxxx | Intent-to-Treat<br>Safety<br>Per-Protocol | xxx | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Population (as ordered above).



# Listing 16.2.4.1: Subject Demographic Information Treatment Arm (Page xx of yy)

| Subject | Eval | B: Date of Birth<br>A: Age<br>S: Sex | R: Race<br>E: Ethnicity | C: Childbearing Potential M: Method of Birth Control | <pre>I: Informed Consent Date P: Photography Consent Signed</pre> |
|---|---|---|---|---|---|
| xxxxx | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxxx | R: xxxxxx xxxxxxx<br>xx xxxxx xxxxxxx<br>xxxxxxx | C: xxx M: xxxxxxxxx xxxxxxxx | I: xxxx-xx-xx<br>P: xxx |
| xxxxxx | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxx | R: xxxxx<br>E: xxxxxxxx xx xxxxxx | C: xx<br>M: | I: xxxx-xx-xx<br>P: xx |
| xxxxx | xxxxxxxx | B: xxxx-xx-xx<br>A: xx<br>S: xxxxxx | R: xxxxx<br>E: xxxxxxxx xx xxxxxx | C: xxx<br>M: xxxxxxxx xxxxxxxxxxxx | I: xxxx-xx-xx<br>P: xx xxxx x xxxxxxxxxx xxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.



#### Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Medical/Surgical History Verbatim Term |
|---|---|---|
| xxxx xxx xxxxxxxx xxxxxx xxxxxxxx | xxxxxxx | xxxxxx |
| | xxxx xxxxxxxx xxxxxxx | xxxx xxxxxxxxx xxxxxx |
| xxxxxxxx xxx xxxxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| | xxxxxxxxxxx | xxxxxxxxxxx x xxxx xxx xxx |
| | | *********** ** ***** ** **** |

Note: System Organ Class and Preferred Term map to MedDRA (Version 21.0).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, and Verbatim Term.



### Listing 16.2.4.2.2: Medical/Surgical History Treatment Arm (Page xx of yy)

| | | | Medical/Surgical History | S: MedDRA System Organ Class | S: Onset Date |
|---|---|---|---|---|---|
| Subject | Age/Sex | Eval | Verbatim Term | P: MedDRA Preferred Term | E: End Date |
| ××××× | xxxx | xxxxxxx | xxxxxx | S: xxxx xxx xxxxxxxxxx xxxxx xxxxx xxxxxx | S: xxxx |
| | | | | P: xxxxxxx | E: |
| | | | ****** ** ******** ******* | S: xxxxxx xxxxxx xxxxxxxxx | S: xxxx |
| | | | | P: xxxxxxx xxxxx xxxxxx | E: xxxxxxx |
| xxxxx | xxxx | xxxxxxx | xxxxxx | S: xxxx xxx xxxxxxxxxx xxxxx xxxxxxx | S: xxxx |
| | | | | P: xxxxxxx | E: |
| xxxxxx | XXXX | xxxxxxxx | xxxxxxx | S: xxxx xxx xxxxxxxxxx xxxxx xxxxxxxx | S: xxxx |
| | | | | P: xxxxxxx | E: |
| xxxxxx | XXXX | xxxxxxxx | xxxxxx | S: xxxx xxx xxxxxxxxxx xxxxxx xxxxxxxx | S: xxxx |
| | | | | P: xxxxxxx | E: |
| | | | xxxxxxxxxxxxx | S: xxxxx xxxxx xxxx | S: xxxxxxxxxx |
| | | | | P: xxxx xxxxxxxxxx | E: xxxxxxxx |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Acne Diagnosis (all Acne MH will appear first), Onset Date, End Date, Verbatim Term



#### Listing 16.2.4.3.1: Unique Medication Names Coded to WHO Drug Global Dictionary ATC Level 2 Terms and Preferred Names (Page xx of yy)

| WHO ATC Level 2 Term | WHO Preferred Name | Medication Verbatim Term | <pre>I: Indication T: Route</pre> |
|---|---|---|---|
| xxxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxx | I: xxxxxxxxxxx<br>R: xxxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |
| xxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | I: xxxxxxxxxxx<br>R: xxxxxxxxxxx |
| | | xxxxxxxx | I: xxxxxxxxxx<br>R: xxxxxxxxxx |

Note: ATC Level 2 Term and Preferred Name map to WHO Drug Global Dictionary, Format B3, Version March 1, 2018

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Preferred Name, Medication Verbatim Term, Indication, and Route.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



### Listing 16.2.4.3.2: Prior and Concomitant Medications Treatment Arm (Page xx of yy)

| S: Subject | A: ATC Level 2 Term | S: Start Date (Day) 1 | I: Indication | |
|---|---|---|---|---|
| A: Age/Sex | P: Preferred Name | E: End Date (Day) 1 | | F: Frequency |
| E: Eval | M: Medication Name | P: Prior/Concomitant | U: Units | T: Route |
| S: xxxxxx | A: xxxxxxxx xxx xxxxxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xxx |
| A: xxxx | P: xxxxxxxxxx xxxxxxx xxxxxxxxx xxx xxxxxx | E: xxxxxxxxxxxxxx | D: xx | T: xxxxxxxxxxxxxx |
| E: xxxxxxxx | M: XXXXXX XXXXX XXXXXXXX | P: xxxxxxxxxxxxxxxxx | x U: xxxxxxxxxx | |
| | A: xxxxxxx xx xxxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xx |
| | P: xxxxxxxxxx xxxxxx xxx | E: xxxxxxxxxxxxxx | D: xx | T: xxxxx |
| | M: xxxxxx xxxxxxxxx | P: xxxxx | U: xxxxxxxx | |
| S: xxxxxx | A: xxxxxxxxx xxx xxxxxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xxx |
| A: xxxx | P: xxxxxxxxx xxxxxx xxxxxxx xxx xxx xxx | E: xxxxxxxxxxxxxx | D: xx | T: xxxxxxxxxxxxxx |
| E: xxxxxxxx | M: xxxxxx xxxxx xxxxxxxxx | P: xxxxxxxxxxxxxxxxx | x U: xxxxxxxxxx | |
| | A: xxxxxxx xx xxxxxxx | S: xxxxxxxxxxxxxx | I: xxxxxxx | F: xx |
| | P: xxxxxxxxxx xxxxxx xxx | E: xxxxxxxxxxxxxx | D: xx | T: xxxxx |
| | M: xxxxx xxxxxxxx | P: xxxxx | U: xxxxxxxx | |

Note: ATC Level 2 Term and Preferred Name map to WHO Drug Global Dictionary, Format B3, Version March 1, 2018

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, Route, Frequency. If the Route is Topical, then the area treated is presented within parenthesis (T: Topical (specify area)).

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



### Listing 16.2.4.4.1: Unique Procedure/Therapy Names Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Procedure/Therapy Verbatim Term | Indication |
|---|---|---|---|
| xxxxxxxxxxxx | xxxxxxxxxxx | xxxxxxxx xx xxxxx | xxxxxxxxxx |
| | | xxxxxxxx | xxxxx xx xxxx |
| xxxxxxxxxxxx | xxxxxxxxxxx | xxxxxxx | xxxxxxx |
| | | | xxxxxxxxx |
| | | xxxxxxxx | xxxxxxxxx |
| xxxxx xxx xx xxxxxxx | xxxxxx xxxxxx xxxx | xxxxxxx xxxxxx | xxxxxxx xxxxxxx xx xx xxxxx |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, Verbatim Term, and Indication.



### Listing 16.2.4.4.2: Prior and Concomitant Procedures/Therapies Treatment Arm (Page xx of yy)

| | | | S: MedDRA System Organ Class P: MedDRA Preferred Term | S: Start Date (Day) <sup>1</sup> E: End Date (Day) <sup>1</sup> | T. Indication |
|---|---|---|---|---|---|
| 2 | 7 / C | Prop 1 | | · | I: Indication |
| Subject<br> | Age/Sex | Eval | M: Procedure/Therapy Name | P: Prior/Concomitant | A: Anatomical Area Treated |
| xxxxx | xxxx | xxxxxxx | S: xxxxxx xxx xxxxxxx xxxxxxx | S: xxxxxxxxxxxxxxxx | I: xxxxx xxxxxxx |
| | | | P: xxxxxxxxxx xxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxxx | A: |
| | | | M: xxxxxxx xxxxx xxxxxxx xxxxxxx | P: xxxxxxxxxxxxxxx | |
| xxxxx | XXXX | xxxxxxx | S: xxxxxxx xxx xxxxxxxx xxxxxxxx | S: xxxxxxxxxxxxxxxx | I: xxxxx xxxxxxx |
| | | | P: xxxxxxxxxx xxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxx | A: |
| | | | M: xxxxxx xxxxx xxxxxx xxxxxx | P: xxxxxxxxxxxxxxxx | |
| xxxxx | XXXX | xxxxxxx | S: xxxxxx xxx xxxxxxx xxxxxxx | S: xxxxxxxxxxxxxxxx | I: xxxxx xxxxxxx |
| | | | P: xxxxxxxxxx xxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxx | A: |
| | | | M: xxxxxxx xxxxx xxxxxx xxxxxx | P: xxxxxxxxxxxxxxxx | |
| | | | S: xxxxxx xxxxxxx xxxx | S: xxxxxxxxxxxxxxxx | I: xxxxxxxx xxxxx xx xx |
| | | | P: xxx xxxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxxx | A: xxxxxxxxx |
| | | | M: xxxxxx xxxxxxx | P: xxxxxxxxxxxxxxx | |
| | | | S: xxxxxx xxxxxxx xxxx | S: xxxxxxxxxxxxxxxx | I: xxxxxxxx xxxxx xx xx |
| | | | P: xxx xxxxxxxxx xxxxxxx | E: xxxxxxxxxxxxxxx | A: xxxxxxxxx |
| | | | M: xxxxxx xxxxxxx | P: xxxxxxxxxxxxxxxx | |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Procedure/Therapy Name, and Indication.

Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



### Listing 16.2.5.1: Study Visit Compliance Treatment Arm (Page xx of yy)

Reason Screening Within And Baseline Visit Occurred on Reason for Study Subject Age/Sex Eval Visit Visit Date  $Day^1$ Window<sup>2</sup> Different Days Unscheduled Visit XXXXXX XXXX XXXXXXXX XXXXXXXX XXXXXXXXX XX XXX XXXXXXX XXXXXXXXX XX XXX XXXXXXX XXX XX XXXXXXXXX XXXX X XXXXXXXXXXXX XXX XXXX X XXXXXXXXX XXX XXXX X XXXXXXXXX XX XXX XXXX XXXXX XXXXXXXXXXXX XXX XXXXXX XXXX XXXXXXXX XXXXXXXX XX XXX XXXXXXXXX XXXXXXX XXXXXXXXX XXX XXXX X XXXXXXXXX XX XXX XXXX X XXXXXXXXX XX XXX XXXXXXXXXX XXXXX XXX XXXXXXXXX XX XXXXXXXXXXXXX XXXXXXXXX XX XXX XXXX XXXXX XXXXXXXXX XX XXX XXXXXX XXXX XXXXXXXX XXXXXXXX XXXXXXXXX XX XXX XXXXXXXXX XXX XXXXXXXX XX XXXX X XXX XXXX XX XXX XXX XXXX XXXX X XXX XXXX XX XXX XXX XXXX XXXX X XXXXXXXXX XX XXX XXXX XXXXX XXXXXXXXX XX XXX

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

<sup>1</sup> Day is calculated as date - Baseline date for dates prior to Baseline visit. Otherwise, day is calculated as date - Baseline date + 1 for dates on or after Baseline visit.

<sup>&</sup>lt;sup>2</sup> Determined by protocol-specified visit window for scheduled visits after Baseline.



### Listing 16.2.5.2: Subject Dosing Compliance Treatment Arm (Page xx of yy)

Maximum Number Number of Calculated1 Amount of of Consecutive Date of First Date of Last Days of Number of Study Drug Missed Percent Subject Age/Sex Eval Application Application Exposure Applications Used (g) Applications Compliant Compliant<sup>2</sup> XXXXXX XXXX XXXXXXX XXXXXXXX XXXXXXXXX XX XX XXXX XX XXXXX XXX XXXXXXXXX XXXXXX XXXX XXXXXXX XXXXXXXX XXXX XXXX XXXXXXX XXXXXXXXX XXXX XXXXXXXX XXXXXXXXX XXXXXXXXX XXXXXX XXXXX XXXxxxxxxXXXX XXXXXXX XXXXXXXX XXXXXXXXX XXXXXXXX XXXXXXX XXXXXXX XXXXXXXX XXXXXXXX XXXXXXXXX XX XXXX XXXXX XXX XXXXXX XX XX

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject.

<sup>&</sup>lt;sup>1</sup> The total number of applicationss was calculated using the date of first application, date of last application, and number of applied applications at a deviation.

<sup>&</sup>lt;sup>2</sup> A subject was considered compliant with the dosing regimen if the subject did not miss more than 5 consecutive days applying and applied 80-120% of expected applications based on the length of their participation in the study.



### Listing 16.2.5.3: Subject Dosing Deviations Treatment Arm (Page xx of yy)

Number of Applications Applied Subject Age/Sex Eval Date of Dosing Deviation (Day) 1 xxxxxx XXXX XXXXXXX XXXXXXXXXXXX Х Х XXXXXXXXXXXX XXXXXX XXXX XXXXXXX XXXXXXXXXXXX Х XXXXXX XXXX XXXXXXXX XXXXXXXXXXXX Х XXXXXXXXXXXX Х XXXXXXXXXXXX Х XXXXXXXXXXXX Х xxxxxxxxxxxx Х XXXXXXXXXXXX Х xxxxxx XXXX xxxxxxx XXXXXXXXXXXX Х XXXXXXXXXXXX Х XXXXXX XXXX XXXXXXX XXXXXXXXXXXX

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Date of Dosing Deviation.

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



# Listing 16.2.5.4: Study Medication Accountability Log Treatment Arm (Page xx of yy)

| | | | Kit | Kit | Pump | Pump Dispensing | | Ret | urn | Amount |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Age/Sex | Eval | Number | Contents | Identifier | Date | Weight (g) | Date | Weight (g) | Used (g) |
| xxxxxx | xxxx | xxxxxxx | xxxx | xxxx | X | xxxxxxxxx | xxxx | xxxxxxxxx | xxxx | xxxx |
| | | | | xxxx | X | xxxxxxxx | XXXX | xxxxxxxxx | XXXX | xxxx |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | | XXXX | х | xxxxxxxxx | xxxx | xxxxxxxxx | XXXX | XXXX |
| | | | XXXX | XXXX | х | xxxxxxxxx | xxxx | xxxxxxxxx | xxxx | XXXX |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXX XXXX | | |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| xxxxx | XXXX | XXXXXXX | XXXX | XXXX | X | xxxxxxxxx | xxxx | xxxxxxxxx | xxxx | XXXX |
| | | | | XXXX | X | XXX XXXX | | | | |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | | XXXX | X | XXXXXXXXX | XXX XXXX | xxxxxxxxx | XXXX | |
| xxxxx | XXXX | xxxxxxx | xxxx | XXXX | Х | xxxxxxxxx | xxxx | xxxxxxxxx | xxxx | XXXX |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXXXXXXXX | XXX XXXX | |
| | | | | XXXX | X | XXXXXXXXX | XXXX | XXXXXXXXX | XXXX | XXXX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Note to progammers: Kit Contents is the treatment the kit contained.



#### Listing 16.2.5.5: Photography Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Were Photographs Taken | Date Taken |
|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxx | xxxxxxxx |
| | | | XXXX X | XXX | XXXXXXXX |
| | | | xxxx x | XX | |
| | | | XXXX X | XXX | xxxxxxxxx |
| | | | xxxx xxxxx | XXX | xxxxxxxxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxx | xxxxxxxx |
| | | | XXXX X | XXX | xxxxxxxxx |
| | | | xxxx x | XXX | xxxxxxxxx |
| | | | xxxx x | XXX | xxxxxxxxx |
| | | | xxxxxxxxxx xxxxx xxx | XXX | xxxxxxxxx |
| | | | xxxx xxxxx | XX | |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxx | xxxxxxxxx |
| | | | xxxx x | XXX | xxxxxxxxx |
| | | | xxxx x | XXX | xxxxxxxxx |
| | | | xxxx x | XXX | xxxxxxxxx |
| | | | xxxx xxxxx | XXX | xxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.6.1: Investigator Global Assessment Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Evaluator<br>Initials | Result |
|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | XXXXXXXXX |
| | | | XXXX XXXXX | XXXXXXXXX | XXX | xxxxxxxxx |
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | XXXX XXXXX | XXXXXXXXX | XXX | xxxxxxxxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx x | xxxxxxxxx | XXX | xxxxxxxxx |
| | | | xxxx xxxxx | xxxxxxxxx | XXX | xxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.6.2: Lesion Counts Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Fval | Visit | Date of<br>Assessment | Evaluator<br>Initials | Total<br>Inflammatory<br>Lesion Count | Nodules/Cysts | Total<br>Non-Inflammator<br>Lesion Count |
|---|---|---|---|---|---|---|---|---|
| | nge/bex | | VISIC | | 111111111111111111111111111111111111111 | Ecsion count | Modules/ cyses | nesion counc |
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxx | xx | XX | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | XX | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | XX | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | xx | xx |
| | | | xxxx xxxxx | xxxxxxxxx | XXX | XX | XX | XX |
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxx | XX | XX | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | xx | xx |
| | | | XXXX X | xxxxxxxxx | XXX | XX | xx | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | xx | xx |
| | | | xxxx xxxxx | xxxxxxxxx | xxx | XX | XX | XX |
| XXXXX | XXXX | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxx | xx | XX | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | XX | XX |
| | | | xxxx x | xxxxxxxxx | XXX | XX | xx | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | XX | XX |
| | | | xxxx xxxxx | xxxxxxxxx | XXX | XX | XX | XX |
| XXXXX | XXXX | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxx | xx | XX | XX |
| | | | XXXX X | xxxxxxxxx | XXX | XX | XX | xx |
| | | | XXXX X | XXXXXXXXX | XXX | XX | XX | XX |
| | | | XXXX XXXXX | XXXXXXXXX | XXX | XX | XX | XX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



#### Listing 16.2.6.3.1: Acne-QoL Descriptions 

| Number | Acne-QoL Question |
|---|---|
| 1 | In the past WEEK, how unattractive did you feel because of your facial acne? |
| 2 | In the past WEEK, how embarrassed did you feel because of your facial acne? |
| 3 | In the past WEEK, how self-conscious (uneasy about oneself) did you feel about your facial acne? |
| 4 | In the past WEEK, how upset were you about having facial acne? |
| 5 | In the past WEEK, how annoyed did you feel at having to spend time every day cleaning and treating your face because of your facial acne? |
| 6 | In the past WEEK, how dissatisfied with your self-appearance did you feel because of your facial acne? |
| 7 | In the past WEEK, how concerned or worried were you about not looking your best because of your facial acne? |
| 3 | In the past WEEK, how concerned or worried were you that your acne medication/products were working fast enough in clearing the acne on your face? |
| 9 | In the past WEEK, how bothered did you feel about the need to always have medication or cover-up available for the acne on your face? |
| 10 | In the past WEEK, how much was your self-confidence (sure of yourself) negatively affected because of your facial acne? |
| 11 | In the past WEEK, how concerned or worried were you about meeting new people because of your facial acne? |
| 12 | In the past WEEK, how concerned or worried were you about going out in public because of your facial acne? |
| 13 | In the past WEEK, how much was socializing with people a problem for you because of your facial acne? |
| 14 | In the past WEEK, how much was interacting with the opposite sex (or same sex if gay or lesbian) a problem for you because of your facial acne? |
| 15 | In the past WEEK, how many bumps did you have on your face? |
| 16 | In the past WEEK, how many bumps full of pus did you have on your face? |

TOOL.AN.10-01.01 Statistical Analysis Plan Template



### Listing 16.2.6.3.1: Acne-QoL Descriptions 

| Number | Acne-QoL Question |
|---|---|
| 17 | In the past WEEK, how much scabbing from your facial acne did you have? |
| 18 | In the past WEEK, how concerned or worried were you about scarring from your facial acne? |
| 19 | In the past WEEK, how oily was your facial skin? |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



## Listing 16.2.6.3.2: Acne-QoL Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | xxxxxxx | xxxxxxxxx<br>xxxxxxxxx | xxxxxxxxx<br>xxxxxxxxx | X<br>X | x<br>x | x<br>x | х | X<br>X | X<br>X | x<br>x | X<br>X | х | X<br>X | х | X<br>X | x<br>x | X<br>X | X<br>X | X<br>X | X<br>X | X<br>X | X<br>X |
| xxxxxx | xxxxx | xxxxxxx | xxxxxxxxx<br>xxxxxxxx | xxxxxxxxx<br>xxxxxxxx | x<br>x | X<br>X | X<br>X | х | X<br>X | X<br>X | X<br>X | x<br>x | X<br>X | X<br>X | Х | X<br>X | X<br>X | x<br>x | X<br>X | X<br>X | Х | X<br>X | x<br>x |
| xxxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | Х | х | Х | Х | х | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | Х | Х | Х | Х |
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | ***** | X | х | x | x | x | x | x | x | x | x | X | х | х | х | x | х | X | X | х |
| | | | XXXXXXXXX | xxxxxxxxx | Х | Х | X | Х | X | X | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | Х | Х | Х |
| XXXXXX | XXXXX | XXXXXXX | xxxxxxxxx<br>xxxxxxxx | XXXXXXXXXX | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Note: Questions 1-14, 18-19: 0=Extremely, 1=Very Much, 2=Quite A Bit, 3=A Good Bit, 4=Somewhat, 5=A Little Bit, 6=Not At All. Questions 15-17: 0=Extensive, 1=A Whole Lot, 2=A Lot, 3=A Moderate Amount, 4=Some, 5=Very Few, 6=None.

ND = NOT DONE

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



# Listing 16.2.6.3.3: Acne-QoL Domain Scores Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Self Perception | Role-social | Role-emotional | Acne Symptoms |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | xx | xx | xx | xx |
| | | | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| | | | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | XX | XX | xx | XX |
| | | | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | XX | XX | xx | XX |
| | | | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| | | | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| | | | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxx | xxxxx | xxxxxxx | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| | | | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| xxxxxx | xxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | XX | XX | XX | XX |
| | | | xxxxxxxxx | xxxxxxxx | xx | XX | xx | XX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



## Listing 16.2.6.4: PRO - Patient Reported Evaluation of Facial Acne (PRE-FACE) Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Category | Assessment | Result |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | Signs/Symptoms | Rate the pimples on your face today | Х |
| | | | | | | Rate the blackheads on your face today | х |
| | | | | | | Rate the whiteheads on your face today | Х |
| | | | | | | Rate the redness on your face today | Х |
| | | | | | Impacts | Over the past seven days, rate how embarrassed you felt because of the acne on your face | Х |
| | | | | | | Over the past seven days, rate how sad you felt because of the acne on your face. | Х |
| | | | xxxx x | xxxxxxxxx | Signs/Symptoms | Rate the pimples on your face today | х |
| | | | | | | Rate the blackheads on your face today | Х |
| | | | | | | Rate the whiteheads on your face today | Х |
| | | | | | | Rate the redness on your face today | Х |
| | | | | | Impacts | Over the past seven days, rate how embarrassed you felt because of the acne on your face | Х |
| | | | | | | Over the past seven days, rate how sad you felt because of the acne on your face. | Х |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject and Visit Number, Category (in order presented on eCRF), and Assessment (in order presented on eCRF).

TOOL.AN.10-01.01 Statistical Analysis Plan Template



Listing 16.2.6.5: PRO - Patient Reported Impression of Symptom Severity (PGI-S)

Treatment Arm

(Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Assessment | Result |
|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | Right now, my acne symptoms are | ****** ** ****** *** |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx xx | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx xx | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx x | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxxx xxxx xxx |
| | | | xxxx xx | xxxxxxxxx | Right now, my acne symptoms are | xxxxxx xx xxxxxx xxxx xxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



Listing 16.2.6.6: PRO - Patient Global Impression of Change (PGI-C), Patient Global Impression of Treatment Satisfaction (PGI-TS),

Patient Global Impression of Treatment Side-Effects (PGI-SE)

Treatment Arm

(Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | PRO Category | Object of<br>Assessment | Result |
|---|---|---|---|---|---|---|---|
| XXXXXX XXXX | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | PGI-C<br>PGI-TS<br>PGI-SE | CHANGE<br>SATISFACTION<br>SIDE-EFFECTS | ************************************** |
| | | | xxxxxxxx | xxxxxxxxx | PGI-C<br>PGI-TS<br>PGI-SE | CHANGE<br>SATISFACTION<br>SIDE-EFFECTS | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | xxxxxxxx | xxxxxxxxx | PGI-C<br>PGI-TS<br>PGI-SE | CHANGE<br>SATISFACTION<br>SIDE-EFFECTS | xxxxxxxxxxxx<br>xxxxxx xxx xxxx<br>xxxxxxxxxx |
| | | | xxxxxxxx | xxxxxxxxx | PGI-C<br>PGI-TS<br>PGI-SE | CHANGE<br>SATISFACTION<br>SIDE-EFFECTS | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxx | xxxx | xxxxxx | xxxxxxxx | xxxxxxxxx | PGI-C<br>PGI-TS<br>PGI-SE | CHANGE<br>SATISFACTION<br>SIDE-EFFECTS | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | xxxxxxxx | xxxxxxxxx | PGI-C<br>PGI-TS<br>PGI-SE | CHANGE<br>SATISFACTION<br>SIDE-EFFECTS | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit Number, and PRO Assessment (in order presented on eCRF).



#### 

| Subject | Age/Sex | Eval | Visit | Date of Assessment | Evaluator<br>Initials | Test | Result |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxx | Erythema | xxxxxxx |
| | | | | | | Scaling | xxx xxxx |
| | | Pigmentatior<br>Dryness | | | Pigmentation | xxxxxxxxxxx | |
| | | | Dryness | xxxxxxxxxx | | | |
| | | | | | | Itching | xxxxxxxxxx |
| | | | | | | Burning | xxxxxxxxxx |
| | | | | | | Stinging | xxxxxxxxx |
| | | | xxxx x | xxxxxxxx xxx | | Erythema | xxxxxxx |
| | | | | | | Scaling | xxx xxxx |
| | | | | | | Pigmentation | xxxxxxxxxx |
| | | | | | | Dryness | XXXXXXXXXX |
| | | | | | | Itching | XXXXXXXXXX |
| | | | | | | Burning | xxxxxxxxx |
| | | | | | | Stinging | XXXXXXXXXX |
| | | | xxxx x | xxxxxxxxx xxx | | Erythema | xxxxxxx |
| | | | | | | Scaling | XXX XXXX |
| | | | | | | Pigmentation | xxxxxxxxxx |
| | | | | | | Dryness | xxxxxxxxx |
| | | | | | | Itching | xxxxxxxxx |
| | | | | | | Burning | XXXXXXXXXX |
| | | | | | | Stinging | XXXXXXXXXX |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit Number, and Test (in order presented on eCRF).



### Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms Treatment Arm (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Application<br>Area | Adverse Event |
|---|---|---|---|
| ******* ******************************* | ******** | xxx | ********** |
| | | xx | xxxxxxx |
| | | xx | xxxxx xxxxxxxx |
| | xxxxxxxx | xx | xxxxxxx |
| ***** | xxxxxxx | xx | xxxxxx |
| **** *** ********* ***** | xxxxxxx | xxx | ****** |
| | xxxx xxxxxxxxxx | xx | xxxxxx xxxx xxxxxxxx xxxx |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, Adverse Event.



### Listing 16.2.7.2.2: Pre-Treatment Adverse Events Treatment Arm (Page xx of yy)

A: In the Application Area S: Subject S: MedDRA System Organ Class G: Severity A: Action Taken with Study Drug A: Age/Sex P: MedDRA Preferred Term R: Relationship to Study Drug T: Action Taken to Treat Event S: Start Date (Day) 1 E: Eval A: Adverse Event S: Serious Event O: Outcome E: End Date (Day) 1 S: xxxxxx S: xxxx xxx xxxxxxxxx xxxxxx A: xx A: xxx xx xxxxxxx S: xxxxxxxxxxxxxxx A: xxxx P: xxx xxxxxxxxxx G: xxxx T: xxxx E: xxxxxxxxxxxxxxx E: xxxxxxx A: xxxxxxx xxxx xxxxxxxx xxxx R: xxx xxxxxxx O: xxxxxxxxxxxxxxxx S: xx S: xxxxxxx xxxxxxxx xxx xxxxxxxx A: xxx A: xxx xxxxxxxxx S: xxxxxxxxxxxxxxx T: xxxxxxxxxxx xxxxxxxx P: xxxxxxxxxx G: xxxx E: xxxxxxxxxxxxxA: xxxxxxxx xxxxx xxxxxx xxxx R: xxx xxxxxxx O: xxxxxxxxxxxxxxxxx S: xx S: xxxxxx S: xxxx xxxxxxxx xxxxx A: xx A: xxx xx xxxxxxx S: xxxxxxxxxxxxxxx A: xxxx P: xxxxxxxxx G: xxxxxxxx T: xxxx E: xxxxxxxxxxxxxx E: xxxxxxxx A: xxxxxxxx xxxxx R: xxx xxxxxxx O: xxxxxxxxxxxxxxxxx S: xx S: xxxxxx S: xxxx xxxxxxxx xxxxxx A: xx A: xxx xx xxxxxx S: xxxxxxxxxxxxxxx A: xxxx P: xxxxxxxxx G: xxxxxxxx T: xxxx E: xxxxxxxxxxxxxxx O: xxxxxxxxxxxxxxxx E: xxxxxxxx A: xxxxxxxx xxxxx R: xxxxxxx S: xxx S: xxxxxxx xxxxxxxx xxx xxxxxxxx A: xxx xxxxxxxxx S: xxxxxxxxxxxxxx A: xxx P: xxxxxxxxxx G: xxxx T: xxxxxxxxxxx xxxxxxxx E: xxxxxxxxxxxxxxx A: xxxxxxxx xxxxx xxxxxxx xxxx R: xxx xxxxxxx O: xxxxxxxxxxxxxxxx S: xx


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Adverse Event.

<sup>1</sup> Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



### Listing 16.2.7.2.3: Treatment-Emergent Adverse Events Treatment Arm (Page xx of yy)

A: In the Application Area S: Subject S: MedDRA System Organ Class G: Severity A: Action Taken with Study Drug A: Age/Sex P: MedDRA Preferred Term R: Relationship to Study Drug T: Action Taken to Treat Event S: Start Date (Day) 1 E: Eval A: Adverse Event S: Serious Event O: Outcome E: End Date (Day) 1 S: xxxxxx S: xxxx xxx xxxxxxxxx xxxxxx A: xx A: xxx xx xxxxxxx S: xxxxxxxxxxxxxxx E: xxxxxxxxxxxxxxx A: xxxx P: xxx xxxxxxxxxx G: xxxx T: xxxx E: xxxxxxx A: xxxxxxx xxxx xxxxxxxx xxxx R: xxx xxxxxx O: xxxxxxxxxxxxxxxx S: xx S: xxxxxxx xxxxxxxx xxx xxxxxxxx A: xxx A: xxx xxxxxxxxx S: xxxxxxxxxxxxxxx T: xxxxxxxxxxx xxxxxxxx P: xxxxxxxxxx G: xxxx E: xxxxxxxxxxxxxA: xxxxxxxx xxxxx xxxxxx xxxx R: xxx xxxxxxx O: xxxxxxxxxxxxxxxxx S: xx S: xxxxxx S: xxxx xxxxxxxx xxxxxx A: xx A: xxx xx xxxxxxx S: xxxxxxxxxxxxxxx A: xxxx P: xxxxxxxxx G: xxxxxxxx T: xxxx E: xxxxxxxxxxxxxx E: xxxxxxxx A: xxxxxxxx xxxxx R: xxx xxxxxxx O: xxxxxxxxxxxxxxxxx S: xxx S: xxxxxx S: xxxx xxxxxxxx xxxxxx A: xx A: xxx xx xxxxxx S: xxxxxxxxxxxxxxx A: xxxx P: xxxxxxxxx G: xxxxxxxx T: xxxx E: xxxxxxxxxxxxxxx O: xxxxxxxxxxxxxxxx E: xxxxxxxx A: xxxxxxxxx xxxxx R: xxx xxxxxxx S: xxx S: xxxxxxx xxxxxxxx xxx xxxxxxxx A: xxx xxxxxxxxx S: xxxxxxxxxxxxxx A: xxx P: xxxxxxxxxx G: xxxx T: xxxxxxxxxxx xxxxxxxx E: xxxxxxxxxxxxxxx R: xxxxxxx A: xxxxxxxx xxxxx xxxxxxx xxxx O: xxxxxxxxxxxxxxxx


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Adverse Event.

<sup>1</sup> Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



### Listing 16.2.7.2.4: Serious Adverse Events Treatment Arm (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | S: MedDRA System Organ Class P: MedDRA Preferred Term A: Adverse Event O: Occurred Prior to First Application | <del>=</del> | A: Action Taken with Study Dru<br>T: Action Taken to Treat Event<br>O: Outcome | = |
|---|---|---|---|---|
| S: xxxxxx | S: xxxx xxx xxxxxxxxxx xxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxx |
| A: xxxx<br>E: xxxxxxxx | P: xxx xxxxxxxxxx<br>A: xxxxxx xxxx xxxxxxxx xxxxx | G: xxxx<br>R: xxx xxxxxxx | T: xxxx O: xxxxxxxxxxxxxxx | E: xxxxxxxxxxxxxx |
| L. AAAAAAAA | 0: xx | S: xxx | U. AAAAAAAAAAAAAAA | |
| | S: xxxxxx xxxxxxx xxx xxxxxxx | A: xxx | A: xxx xxxxxxxxx | S: xxxxxxxxxxxxx |
| | P: xxxxxxxxx | G: xxxx | T: xxxxxxxxxxx xxxxxxxx | E: xxxxxxxxxxxxxx |
| | A: xxxxxxxx xxxxx xxxxxx xxxx<br>O: xx | R: xxx xxxxxxx<br>S: xxx | 0: xxxxxxxxxxxxxxx | |
| S: xxxxxx | S: xxxx xxxxxxxx xxxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxxx |
| A: xxxx | P: xxxxxxxx | G: xxxxxxxx | T: xxxx | E: xxxxxxxxxxxxxx |
| E: xxxxxxxx | A: xxxxxxxx xxxxx | R: xxxxxxx | O: xxxxxxxxxxxxxxxx | |
| | 0: xx | S: xxx | | |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Adverse Event.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

<sup>1</sup> Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



Listing 16.2.7.2.5: Subjects Who Prematurely Discontinued Study and/or Discontinued Study Drug Due to Adverse Events

Treatment Arm

(Page xx of yy)

| | S: MedDRA System Organ Class | | | |
|---|---|---|---|---|
| | P: MedDRA Preferred Term | A: In the Application Area | | |
| S: Subject | A: Adverse Event | G: Severity | A: Action Taken with Study Dru | ıg |
| A: Age/Sex | O: Occurred Prior to First | R: Relationship to Study Drug | T: Action Taken to Treat Event | S: Start Date (Day) |
| E: Eval | Application | S: Serious Event | O: Outcome | E: End Date (Day) 1 |
| S: xxxxxx | S: xxxx xxx xxxxxxxxxx xxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxxx |
| A: xxxx | P: xxx xxxxxxxxxx | G: xxxx | T: xxxx | E: xxxxxxxxxxxxxx |
| E: xxxxxxxx | A: xxxxxxx xxxx xxxxxxxx xxxxx | R: xxx xxxxxxx | O: xxxxxxxxxxxxxxxx | |
| | O: xx | S: xxx | | |
| | S: xxxxxx xxxxxxxx xxx xxxxxxxx | A: xxx | A: xxx xxxxxxxxx | S: xxxxxxxxxxxxxx |
| | P: xxxxxxxxxx | G: xxxx | T: xxxxxxxxxxx xxxxxxxx | E: xxxxxxxxxxxxxx |
| | A: xxxxxxxx xxxxx xxxxxxx xxxx | R: xxx xxxxxxx | O: xxxxxxxxxxxxxxxx | |
| | O: xx | S: xxx | | |
| S: xxxxxx | S: xxxx xxxxxxxx xxxxxx | A: xx | A: xxx xx xxxxxxx | S: xxxxxxxxxxxxxx |
| A: xxxx | P: xxxxxxxxx | G: xxxxxxxx | T: xxxx | E: xxxxxxxxxxxxxx |
| E: xxxxxxxx | A: xxxxxxxx xxxxx | R: xxxxxxx | 0: xxxxxxxxxxxxxx | |
| | 0: xx | S: xxx | | |


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Adverse Event.

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first application for dates prior to first application. Otherwise, day is calculated as date - date of first application + 1 for dates on or after first application.



# Listing 16.2.8.1: Urine Pregnancy Tests Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of Assessment | Results | Reason Test Not Done |
|---|---|---|---|---|---|---|
| XXXXXX | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxx | |
| | | | XXXXXXX | XXXXXXXXX | XXXXXXXX | |
| | | | XXXX X | | | XXX XXXX |
| | | | XXXX X | XXXXXXXXX | XXXXXXXX | |
| | | | XXXX X | xxxxxxxxx | XXXXXXX | |
| XXX | XXXX | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxx | |
| | | | xxxxxxxx | xxxxxxxxx | XXXXXXXX | |
| | | | xxxx x | xxxxxxxxx | XXXXXXXX | |
| | | | xxxx x | xxxxxxxxx | XXXXXXXX | |
| | | | XXXX X | xxxxxxxx | XXXXXXX | |
| XXX | XXXX | xxxxxxxx | xxxxxxxxx | | | xxx xxxxxxxxx |
| | | | xxxxxxxxx | | | XXX XXXXXXXXX |
| | | | xxxx x | | | xxx xxxxxxxxx |
| | | | xxxx x | | | xxx xxxxxxxxx |
| | | | xxxx x | | | xxx xxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)



## Listing 16.2.8.2: Physical Examination Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Body System | Exam Finding | Reason Exam<br>Not Done |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | xxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxx<br>xxxx<br>xxxxxxx<br>xxxxxxxxxxxxxxxxxxx | ******* ******* ******* ******* **** | |
| | | | XXXX XXXXX | xxxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxx xxxx<br>xxx xxxx | *** ********************************** |
| xxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | xxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX<br>XXXXXXX<br>XXXXXXXX XXXXXXXXX XXXX<br>XXXXXXX XXXXX XXXX | |
| | | | xxxx xxxxx | xxxxxxxxx | xxxxx<br>xxxxxxxxx<br>xxxxxxxxxxxx<br>xxxxxxxxx | xxx xxxx<br>xxx xxxx<br>xxx xxxx | xxx xxxxxxxxx<br>xxx xxxxxxxxx |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit Number, and Body System (in order presented on eCRF).



# Listing 16.2.8.3: Vital Signs Treatment Arm (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | Vital Sign | Result | Units |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | ******* | xx | xxxx |
| | | | | | XXXXX XXXX | XX | xxxxxxxx |
| | | | | | XXXXXX | xxxxx | xx |
| | | | | | xxxxxxxxxx xxxx | xx | xxxxxxxxxx |
| | | | | | xxxxxxx xxxxx xxxxxxx | xxx | xxxx |
| | | | | | xxxxxxxxxx | xxxx | x |
| | | | | | xxxxxx | XXX | XX |
| | | | xxxx xxxxx | xxxxxxxxx | ****** | XX | xxxx |
| | | | | | XXXXX XXXX | xxx xxxx | |
| | | | | | xxxxxxxxxx xxxx | xxx | xxxxxxxxxx |
| | | | | | XXXXXXX XXXXX XXXXXXX | xxx | xxxx |
| | | | | | xxxxxxxxx | XX | X |
| xxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxxxxxx | ****** | XX | xxxx |
| | | | | | xxxxx xxxx | xx | xxxxxxxxx |
| | | | | | xxxxxx | xxx | XX |
| | | | | | xxxxxxxxxx xxxx | XX | xxxxxxxxxx |
| | | | | | xxxxxxx xxxxx xxxxxxx | XX | xxxx |
| | | | | | XXXXXXXXX | XX | Х |
| | | | | | xxxxxx | XXX | XX |
| | | | xxxx xxxxx | xxxxxxxxx | xxxxxxxx xxxxx xxxxxxx | xxx xxxx | |
| | | | | | xxxxx xxxx | xxx xxxx | |
| | | | | | xxxxxxxxxx xxxx | xxx xxxx | |
| | | | | | xxxxxxx xxxxx xxxxxxx | xxx xxxx | |
| | | | | | xxxxxxxxxx | xxx xxxx | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit Number, and Vital Sign (in alphabetical order).